

Innovation for patient care

D-CN-52014-237


# PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024

#### **Protocol Title:**

A multicentre, open-label, single-arm study to investigate the efficacy and safety of triptorelin pamoate 22.5 mg 6-month formulation in Chinese patients with locally advanced or metastatic prostate cancer

Protocol Number: D-CN-52014-237

**Compound:** Triptorelin pamoate (embonate) salt (IPN52014)

**Short Title:** Effects of triptorelin pamoate 6-month when given to adult Chinese participants with advanced cancer in the prostate

Study Phase: IIIb

**Sponsor Name:** Ipsen Pharma

## **Legal Registered Address:**

Ipsen Pharma 65, quai Georges Gorse 92100 Boulogne Billancourt, France

#### **Regulatory Authority Identifier Number(s)**

Not applicable

**Date:** 08 March 2024

Version Number: 4.0 Amendment Number: 3

Persons supplied with this information must understand that it is strictly confidential.

Information contained herein cannot be disclosed, submitted for publication or used for any purpose other than that contemplated herein without the sponsor's prior written authorisation.

Date

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 2/92

# Sponsor Signatory:

PPD

Medical Development Director

R&D Shanghai Innovation Hub Ipsen (Shanghai)

Unit 01, 15th Floor

No.218, Xujiahui Road

Huangpu District

Shanghai 200001

China

#### Medical Monitor Name and Contact Information:

PPD

Medical Development Director

R&D Shanghai Innovation Hub Ipsen (Shanghai)

Unit 01, 15th Floor

No.218, Xujiahui Road

Huangpu District

Shanghai 200001

China

Telephone: PPD

IPSEN GROUP D-CN-52014-237


PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 3/92

### **Principal Investigator Signature Page**

I have read and agree to Protocol D-CN-52014-237 entitled "A multicentre, open-label, single-arm study to investigate the efficacy and safety of triptorelin pamoate 22.5 mg 6-month formulation in Chinese patients with locally advanced or metastatic prostate cancer" with protocol Amendment #3. I am aware of my responsibilities as an investigator under the guidelines of Good Clinical Practice (GCP), local regulations (as applicable) and the study protocol. I agree to conduct the study according to these guidelines and to appropriately direct and assist the staff under my control, who will be involved in the study.

| NAME: | (l) | |
|---------|--------------|------------|
| TITLE: | [PRINCIPAL] | SIGNATURE: |
| | INVESTIGATOR | |
| DATE: | | |
| OFFICE. | rlh | |
| OFFICE: | [i] | |
| | (l) | |
| | [1] | |


### PROTOCOL AMENDMENT SUMMARY OF CHANGES

| DOCUMENT HISTORY | | | |
|-------------------|---------|------------------|------------|
| Document | Version | Date | Status |
| Amendment 3 | 4.0 | 08 March 2024 | Effective |
| Amendment 2 | 3.0 | 07 April 2022 | Superseded |
| Amendment 1 | 2.0 | 11 November 2021 | Superseded |
| Original Protocol | 1.0 | 31 July 2019 | Superseded |

# Amendment 3 (08 March 2024)

# **Overall Rationale for the Amendment:**

Protocol was updated to clarify ambiguous wording/text in the protocol and the safety/full analysis set.

# Summary change table from previous version of the protocol

Any new or amended text in the protocol is indicated in bold. Deletions are marked in strikeout text. Minor formatting and editing are not included.

| T III. |
|--------|

| Section | Was (Version 3.0, 07 April 2022) | Is (Version 4.0, 08 March 2024) | Rationale |
|---|---|---|---|
| Sponsor<br>Signatory and<br>Medical<br>Monitor Name<br>and Contact<br>Information<br>Page | Sponsor Signatory: PPD Medical Development Director R&D Shanghai Innovation Hub Ipsen (Shanghai) No. 2306 International Capital Plaza No. 1318 North Sichuan Road Shanghai 200080 China Medical Monitor Name and Contact Information: PPD Medical Development Director R&D Shanghai Innovation Hub Ipsen (Shanghai) No. 2306 International Capital Plaza No. 1318 North Sichuan Road Shanghai 200080 China Telephone: PPD | Sponsor Signatory: PPD Medical Development Director R&D Shanghai Innovation Hub Ipsen (Shanghai) Unit 01, 15th Floor No.218, Xujiahui Road Huangpu District Shanghai 200001 China Medical Monitor Name and Contact Information: PPD Medical Development Director R&D Shanghai Innovation Hub Ipsen (Shanghai) Unit 01, 15th Floor No.218, Xujiahui Road Huangpu District Shanghai 200001 China Telephone: PPD | Change of sponsor personnel. |
| 1.3 Schedule of<br>Activities<br>(Table 1 and<br>Table 2) | Footnote "d" Table 1 and Footnote "e" Table 2:<br>Injection site to be specifically checked 2 hours after<br>injection for local reactions on Day 1. After Day 1<br>any local reaction AEs to be collected on the CRF in<br>the same manner as other AEs. | Footnote "d" Table 1 and Footnote "e" Table 2: Injection site to be specifically checked 2 hours ±15 minutes after injection for local reactions on Day 1. After Day 1 any local reaction AEs to be collected on the CRF in the same manner as other AEs. | Reasonable time window is allowed for applicability. |


| Section | Was (Version 3.0, 07 April 2022) | Is (Version 4.0, 08 March 2024) | Rationale |
|---|---|---|---|
| Section 1.3 Schedule of Activities (Table 2) | Was (Version 3.0, 07 April 2022) Footnote "c": Sampling on Day 1. PK time sampling windows: • Pre-dose (≤30 mins) prior to study drug injection • 1h, 2h, 3h post-dose ±5 mins • 4h, 6h, 8h post-dose ±15 mins • 12h post-dose ±30 mins • 24h post-dose ±1 hour • 48h post-dose ±2 hours • 120h post-dose ±3 hours • 168h post-dose ±4 hours • Day 15 (2 weeks post-dose) ±24 hours • Day 22 (3 weeks post-dose) ±24 hours • Day 29, 57, 85, 113, 141, 169 = clinic visit time | Is (Version 4.0, 08 March 2024) Footnote "c": Sampling on Day 1. PK time sampling windows: • Pre-dose (≤30 mins) prior to study drug injection • 1h, 2h, 3h post-dose ±5 mins • 4h, 6h, 8h post-dose ±15 mins • 12h post-dose ±30 mins • 24h post-dose ±1 hour • 48h post-dose ±2 hours • 96h post-dose ±3 hours • 168h post-dose ±4 hours • Day 15 (2 weeks post-dose) ±24 hours | Typo correction. |
| 5.2 Exclusion<br>Criteria | Day 29, 57, 85, 113, 141, 169 = clinic visit time windows (±3 days) 3. Previous history of QT prolongation or concomitant use of medicinal products known to prolong the QT interval or with a known risk of torsades de pointes as per Pharmacovigilance Risk Assessment Committee (PRAC) recommendations. | <ul> <li>Day 15 (2 weeks post-dose) ±24 hours</li> <li>Day 22 (3 weeks post-dose) ±24 hours</li> <li>Day 29, 57, 85, 113, 141, 169 = clinic visit time windows (±3 days)</li> <li>3a. Previous history of QT prolongation or concomitant use of medicinal products known to prolong the QT interval or with a known risk of torsades de pointes</li> </ul> | The label of the used medicinal products will be referred per clinical practice. |
| 5.2 Exclusion<br>Criteria | 4. Metastatic hormone-sensitive prostate cancer with high tumour burden. | 4a. Metastatic hormone-sensitive prostate cancer with high tumour burden. (Note: high tumour burden: presence of visceral metastases and/or at least four bone lesions with at least one lesion outside the vertebral column and/or pelvis per CHAARTED study (Kyriakopoulos 2018). | Definition of high tumour burden added for clarification. |


| Section | Was (Version 3.0, 07 April 2022) | Is (Version 4.0, 08 March 2024) | Rationale |
|---|---|---|---|
| 5.2 Exclusion<br>Criteria | 7. Previous hormone therapy (including abiraterone) for prostate cancer within 6 months prior to study start. 8. Previous cytotoxic chemotherapy treatment within 6 months prior to study start. 9. Use of finasteride or dutasteride within 2 months prior to study start. 14. Participation in another study with an investigational drug or treatment within 3 months prior to study entry or within 5 drug half-lives of the investigational drug (whichever is the longer). | 7a. Previous hormone therapy (including abiraterone) for prostate cancer within 6 months prior to study screening. 8a. Previous cytotoxic chemotherapy treatment within 6 months prior to study screening. 9a. Use of finasteride or dutasteride within 2 months prior to study screening. 14a. Participation in another study with an investigational drug or treatment within 3 months prior to study screening or within 5 drug half-lives of the investigational drug (whichever is the longer). | Clarification of exclusion criteria for consistency within the protocol. |
| 5.2 Exclusion<br>Criteria | 11. Any current use or use within 6 months prior to treatment start of medications which are known to affect the metabolism and/or secretion of androgenic hormones: ketoconazole, aminoglutethimide, oestrogens and antiandrogens. | 11a. Any current use or use within 6 months prior to treatment start of medications which are known to affect the metabolism and/or secretion of androgenic hormones: ketoconazole, aminoglutethimide, oestrogens and antiandrogens. Note: antiandrogen: enzalutamide, apalutamide or darolutamide is allowed (if required per investigator's clinical judgement) due to no interference on the metabolism and/or secretion of androgenic hormones. | Clarification added to allow new generation androgen receptor inhibitors considering as they are not anticipated to affect the metabolism and/or secretion of androgenic hormones. |
| 5.2 Exclusion<br>Criteria | 12. Systemic or inhaled corticosteroids (topical application permitted). | 12a. Current use of systemic or inhaled corticosteroids (topical application permitted). | Clarification of corticosteroid use during the study. |
| 6.2 Preparation,<br>Handling,<br>Storage and | The reconstitution needle should then be changed, and the injection needle (20 G, with safety device) used to administer the product. | The reconstitution needle should then be changed, and the injection needle (20 G, without safety device) used to administer the product. | Typo correction. |

Accountability


| Section | Was (Version 3.0, 07 April 2022) | Is (Version 4.0, 08 March 2024) | Rationale |
|---|---|---|---|
| 7.2 Participant<br>Discontinuation/<br>Withdrawal<br>from the Study | | • A participant will be withdrawn from the study if they have inadequate testosterone suppression (defined as >50 ng/dL detected at least 30 days after administration of study intervention and on two consecutive measurements at least 2 weeks apart, at either a scheduled or unscheduled study visit). | Clarification added to provide guidance for participants who have lack of efficacy during the study. |
| 8.3.2 Vital<br>Signs | Blood pressure, temperature, respiratory rate and heart rate will be assessed as outlined in the SoA (Section 1.3) with an automated device so that measurements are independent of the observer. Blood pressure and heart rate will be recorded after 5 minutes rest in supine position. | Blood pressure, temperature, respiratory rate and heart rate will be assessed as outlined in the SoA (Section 1.3) with an automated device (if possible) so that measurements are independent of the observer. Blood pressure and heart rate will be recorded after 5 minutes rest in supine or seated position. | Clarification added to allow flexibility for respiratory rate and position for blood pressure and heart rate per clinical practice. |
| 8.3.4 Magnetic<br>Resonance<br>Imaging Scan | A magnetic resonance imaging (MRI) scan for prostate gland or the whole body (only if necessary, based on investigator's judgement) will be performed as described in the SoA (Table 1 and Table 2) to confirm disease stage prior to study entry. | A magnetic resonance imaging (MRI) scan for prostate gland or the whole body, only if necessary (based on investigator's judgement), will be performed as described in the SoA (Table 1 and Table 2) to confirm disease stage prior to study entry. | Clarification for consistency with SoA Table 1 and Table 2 footnote "g" and "h", respectively. |
| 9.3 Analysis<br>Sets | Safety Set: The safety set will contain all participants who receive at least one dose of study intervention. Full Analysis Set: All treated participants having at | Safety Set: The safety set will contain all participants who receive the single dose of study intervention. Full Analysis Set: The FAS will contain all | Clarification of the safety and full analysis sets. |
| | least one baseline and at least one post baseline assessment of the primary efficacy endpoint. | treated participants who complete the study or is a treatment failure. | |
| | | Completing the study is defined as having serum testosterone measurement at baseline, | |
| | | Day 29 and Day 169. Treatment failure is | |
| | | defined as escaping castration (testosterone | |
| | | level ≥50 ng/dL) at any assessments on and after Day 29 during the study, or premature discontinuation from the intervention period | |


| Section | Was (Version 3.0, 07 April 2022) | Is (Version 4.0, 08 March 2024) | Rationale |
|---|---|---|---|
| | | due to drug-related reasons (adverse event or death). | |
| 10.1.5<br>Dissemination<br>of Clinical<br>Study Data | • Protocol and result summary will be made publicly available on the US Clinical Trials Registry (ClinicalTrials.gov) and for studies run in the EU/EEA on the EU Clinical Trials Register (www.elinicaltrialsregister.eu). The sponsor also provides clinical trial information to other national clinical trial registries or databases according to local requirements/legislation. | • Protocol and result summary will be made publicly available on the US Clinical Trials Registry (ClinicalTrials.gov). The sponsor also provides clinical trial information to other national clinical trial registries or databases according to local requirements/legislation. | Clarification for studies conducted in China. |

# Other documents impacted:

| Informed consent form | Yes 🛛 No 🗌 |
|---------------------------------|------------|
| Case report form (CRF) | Yes 🛛 No 🗌 |
| Statistical analysis plan (SAP) | Yes 🗌 No 🔀 |

# **TABLE OF CONTENTS**

| PRO | ROTOCOL AMENDMENT SUMMARY OF CHANGES | 4 |
|---|---|---|
| TAI | ABLE OF CONTENTS | 10 |
| LIS | ST OF ABBREVIATIONS | 14 |
| 1 | PROTOCOL SUMMARY | 16 |
| 1.1 | Synopsis | 16 |
| 1.2 | Schema | 19 |
| 1.3 | Schedule of Activities (SoA) | 20 |
| 2 | INTRODUCTION | 25 |
| 2.1 | Study Rationale | 25 |
| 2.2 | Background | 25 |
| 2.3 | Benefit/Risk Assessment | 27 |
| | 2.3.1 Risk Assessment | 27 |
| | 2.3.2 Benefit Assessment | 27 |
| | 2.3.3 Overall Benefit: Risk Conclusion | 28 |
| 3 | OBJECTIVES AND ENDPOINTS | 29 |
| 4 | STUDY DESIGN | 31 |
| 4.1 | Overall Design | 31 |
| 4.2 | Scientific Rationale for Study Design | 31 |
| 4.3 | Justification for Dose | 32 |
| 4.4 | End of Study Definition | 32 |
| 5 | STUDY POPULATION | 33 |
| <b>5.1</b> | Inclusion Criteria | 33 |
| <b>5.2</b> | Exclusion Criteria | 33 |
| 5.3 | 3 Lifestyle Considerations | 34 |
| <b>5.4</b> | Screen Failures | 34 |
| 6 | STUDY INTERVENTION AND CONCOMITANT THERAPY | 35 |
| 6.1 | Study Intervention(s) Administered | 35 |
| <b>6.2</b> | Preparation, Handling, Storage and Accountability | 35 |
| 6.3 | Measures to Minimize Bias: Randomisation and Blinding | 36 |
| | 6.3.1 Randomisation | 36 |
| | 6.3.2 Maintenance of Blinding | 36 |
| 6.4 | Study Intervention Compliance | 36 |
| 6.5 | Dose Modification | 36 |
| 6.6 | Continued Access to Study Intervention after the End of the Study | <i>7</i> 36 |
| <b>6.7</b> | Treatment of Overdose | 36 |
| 6.8 | Concomitant Therapy | 37 |
| 7 | DISCONTINUATION OF STUDY INTERVENTION AND PA | ARTICIPANT |
| | DISCONTINUATION/WITHDRAWAL | |
| <b>7.1</b> | Discontinuation of Study Intervention | 39 |

| | 7.1.1 | Temporary Discontinuation | 39 |
|---|---|---|---|
| 7.2 | | cipant Discontinuation/Withdrawal from the Study39 | |
| 7.3 | Lost to Follow-up | | |
| 8 | | ASSESSMENTS AND PROCEDURES | |
| 8.1 | | aphy | |
| 8.2 | U | Assessments | |
| J | 8.2.1 | Testosterone. | |
| | 8.2.2 | Prostate-specific Antigen | |
| 8.3 | | ssessments | |
| | 8.3.1 | Physical Examinations | |
| | 8.3.2 | Vital Signs | |
| | 8.3.3 | Electrocardiograms | |
| | 8.3.4 | Magnetic Resonance Imaging Scan | |
| | 8.3.5 | Clinical Safety Laboratory Assessments | |
| | 8.3.6 | Local Tolerance | |
| 8.4 | Adverse | Events (AEs) and Serious Adverse Events (SAEs), and Other Safe | |
| | | ıg | • |
| | <i>8.4.1</i> | Time Period and Frequency for Collecting AE and SAE Information | 44 |
| | <i>8.4.2</i> | Method of Detecting AEs and SAEs | 44 |
| | <i>8.4.3</i> | Follow-up of AEs and SAEs | 44 |
| | <i>8.4.4</i> | Regulatory Reporting Requirements for SAEs | 44 |
| | <i>8.4.5</i> | Pregnancy | 44 |
| | 8.4.6 | Disease-Related Events and/or Disease-Related Outcomes N<br>Qualifying as AEs or SAEs | |
| | <b>8.4.</b> 7 | Adverse Events of Special Interest | 45 |
| | <i>8.4.8</i> | Reporting of Study Intervention Errors Including Misuse/Abuse | 45 |
| 8.5 | Pharma | cokinetics | 45 |
| 9 | STATIS | TICAL CONSIDERATIONS | 47 |
| 9.1 | Statistica | al Hypotheses | 47 |
| 9.2 | Sample S | Size Determination | 47 |
| 9.3 | Analysis | Sets | 47 |
| 9.4 | Statistica | al Analyses | 48 |
| | <i>9.4.1</i> | General Considerations | 48 |
| | 9.4.1.1 | Reasons for Exclusion from the Analyses | 48 |
| | 9.4.1.2 | Significance Testing and Estimations | 48 |
| | 9.4.1.3 | Statistical/Analytical Methods | 48 |
| | 9.4.2 | Analysis of Primary Endpoints | 49 |
| | 9.4.3 | Analysis of Secondary Endpoints | 49 |
| | 9.4.3.1 | Prostate-Specific Antigen | 49 |
| | 9.4.3.2 | Pharmacokinetic and Pharmacodynamic Data Analysis | 49 |
| | 9.4.4 | Analysis of Exploratory Endpoint | 50 |

|----------------------|-----------------------------------------|
| PROTOCOL: FINAL with | Amendment 3: Version 4.0, 08 March 2024 |

| PRO | TOCOL | L: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAC | GE 12/92 |
|---|---|---|---|
| | 9.4.4. | .1 Pharmacokinetic/Pharmacodynamic Relationship | 50 |
| | 9.4.5 | • | |
| | 9.4.6 | Subgroups Analyses | 51 |
| | 9.4.7 | | |
| 9.5 | Inter | im Analyses | |
| 10 | | PORTING DOCUMENTATION AND OPERATION ISIDERATIONS | |
| 10.1 | | endix: Regulatory, Ethical, and Study Oversight Considerations | |
| 10.1 | 10.1. | | |
| | 10.1.2 | • | |
| | 10.1.2 | | |
| | 10.1. | | |
| | 10.1. | | |
| | 10.1. | · | |
| | 10.1. | <u> </u> | |
| | 10.1. | | |
| | 10.1.6 | • | |
| 10.2 | | 9 Publication Policyendix: Clinical Laboratory Tests | |
| | | • | |
| 10.3 | | endix: AEs and SAEs: Definitions and Procedures for Recording, Evaluatory, and Reporting | |
| | 10.3. | 1 Definition of AE | 58 |
| | 10.3.2 | 2 Definition of SAE | 59 |
| | 10.3. | 3 Recording and Follow-Up of AE and/or SAE | 60 |
| | 10.3.4 | | |
| 10.4 | | endix: American Joint Committee on Cancer (AJCC) TNM Staging Sys | stem |
| 10.5 | | endix: ECOG Performance Scale | |
| | | endix: Protocol Amendment History | |
| 10.0 | 10.6. | | |
| | 10.6.2 | | |
| 11 | | ERENCES | |
| 11 | KET | EREICES | ······ |
| | | LIST OF TABLES | |
| Tabl | le 1 | Schedule of Activities for All Participants Except | the |
| | | Pharmacokinetic/Pharmacodynamic Subset | 21 |
| Tabl | le 2 | Schedule of Assessments for the Pharmacokinetic/Pharmacodyna<br>Subset of Participants | |
| Tabl | le 3 | Study Risk Assessment | 27 |
| Tabl | le 4 | Objectives and Endpoints | 29 |
| Tabl | le 5 | Study intervention administered | 35 |

| IPSEN GR | OUP | D-CN-52014-237 |
|---|---|---|
| PROTOCO | DL: FINAL with Amendment 3: Version 4.0, 08 March 2024 | PAGE 13/92 |
| Table 6 | Protocol-Required Safety Laboratory Tests | 57 |
| | LIST OF FIGURES | |
| Figure 1 | Study Schema | 19 |

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 14/92

#### LIST OF ABBREVIATIONS

ABBREVIATION Wording Definition

**ADT** Androgen deprivation therapy

**AE** Adverse event

ALT Alanine aminotransferase
AST Aspartate aminotransferase

**AUC** Area under the concentration versus time curve

CA Competent authority
CI Confidence interval

C<sub>max</sub> Maximum concentration

**CRF/eCRF** Case report form/electronic case report form

CFR Code of Federal Regulations
COVID-19 Coronavirus disease 2019

**CRO** Contract research organisation

CSR Clinical study report ECG Electrocardiogram

**EDC** Electronic data capture

**ECOG** Eastern Cooperative Oncology Group

**FAS** Full analysis set

FDA Food and Drug Administration
FSH Follicle-stimulating hormone

**GCP** Good clinical practice

**GnRH** Gonadotropin-releasing hormone

Hb Haemoglobin

**ICF** Informed consent form

**ICH** International Conference on Harmonisation

**IEC** Independent Ethics Committee

i.m. Intramuscular

IMP Investigational Medicinal Product

**IRB** Institutional Review Board

IVF In vitro fertilisation
ITT Intention-to-treat

LC-MS/MS Liquid chromatography tandem mass spectrometry

LH Luteinising hormone

# IPSEN GROUP D-CN-52014-237


PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024


**ABBREVIATION** Wording Definition

**LHRH** Luteinising hormone-releasing hormone

MedDRA Medical Dictionary for Regulatory Activities

NCA Non-compartmental analysis

NCI-CTCAE National Cancer Institute – Common Toxicity Criteria for Adverse

**Events** 

**NOS** Not otherwise specified

PD Pharmacodynamics
PK Pharmacokinetics

PLGA Poly(1actide-CO-glycolide)

PP Per Protocol

**PRAC** Pharmacovigilance Risk Assessment Committee

**PSA** Prostate specific antigen

PT Preferred term

SAE Serious adverse event

SAS® Statistical Analysis Software

SD Standard deviation
SOC System Organ Class

**SOP** Standard Operating Procedure

SUSAR Suspected unexpected serious adverse reactions

**TEAE** Treatment-emergent adverse event

t<sub>cast</sub> Time to castration

t<sub>max</sub> Time to peak serum/plasma concentration

TNM Tumour, lymph nodes, metastases

ULN Upper limit of normal

US United States of America

WBC White blood cells

WHO World Health Organisation

**WHODRUG** WHO Drug Dictionary

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 16/92

#### 1 PROTOCOL SUMMARY

#### 1.1 Synopsis

#### **Protocol Title:**

A multicentre, open-label, single-arm study to investigate the efficacy and safety of triptorelin pamoate 22.5 mg 6-month formulation in Chinese patients with locally advanced or metastatic prostate cancer

#### **Short Title:**

Effects of triptorelin pamoate 6-month when given to adult Chinese participants with advanced cancer in the prostate

#### Rationale:

The 6-month triptorelin formulation (22.5 mg) has been evaluated in a multicentre, non-comparative Phase III study in participants with advanced prostate cancer, conducted between July 2006 and August 2007 [Lundstrom 2009]. The results from the study have shown that the new triptorelin 6-month formulation (22.5 mg) rapidly induces and maintains castration in participants with locally advanced or metastatic prostate cancer. In the intention-to-treat (ITT) population, 97.5% (117/120) of participants were castrated (testosterone level <50 ng/dL) on Day 29, and 93.0% (107/115) of participants maintained castration from Week 8 (Day 57) to end of Week 48. The efficacy results of the 6-month formulation have been reviewed with those obtained in previous studies with the marketed triptorelin 1- and 3-month formulations. Results show that the rate of castration achieved with the 6-month formulation on Day 29, after the first triptorelin injection, was comparable to those with the 1-month and 3-month formulations [Breul 2017].

In terms of local tolerance at the injection site, intramuscular triptorelin injections were well tolerated as confirmed in the phase III study where injection site reactions were assessed by active questioning: 6.7% participants with injection-site reactions reported as adverse events (AEs), which is lower than for other 6-month gonadotropin-releasing hormone (GnRH) formulations [Lundstrom 2009]. In a pooled analysis, very few (<5%) local adverse reactions at the injection site have been reported in clinical studies with all triptorelin sustained-release formulations (1-, 3- and 6 month) [Breul 2017].

The advantage of the sustained-release 6-month triptorelin pamoate formulation is that the reduced frequency of injections will provide greater convenience to both the participants and the physician and it may also improve the participant acceptability and compliance with the injection schedule.

The present study will assess the efficacy and safety of the sustained-release 6-month triptorelin pamoate formulation in Chinese participants with locally advanced or metastatic prostate cancer for confirming the registration of this product in China. At the same time, triptorelin pharmacokinetics (PK) and testosterone pharmacodynamics (PD) will be assessed in in this study population.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 17/92

## Objectives and Endpoints:

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the efficacy of triptorelin pamoate 22.5 mg 6-month formulation in achieving castrate levels of testosterone To evaluate the efficacy of triptorelin pamoate 22.5 mg 6-month formulation in maintaining the castrate levels of serum testosterone | Percentage of participants achieving castrate levels of serum testosterone (<50 ng/dL or 1.735 nmol/L) on Day 29 Percentage of participants maintaining the castrate levels from Week 8 to Week 24 |
| Secondary | |
| To assess the safety profile including local tolerability of triptorelin pamoate 22.5 mg 6-month formulation | <ul> <li>Incidence of TEAEs (including local tolerability) throughout the study i.e., up to Week 24</li> <li>Change from baseline in clinical safety laboratory parameters (blood chemistry and haematology) at Week 24</li> <li>Change from baseline in physical examination at Day 1, Week 12 and Week 24</li> <li>Change from baseline in ECG at Week 4 and Week 24</li> <li>Change from baseline in vital signs (blood pressure and heart rate) at each visit up to Week 24</li> </ul> |
| To demonstrate the effect of triptorelin<br>pamoate 22.5 mg 6-month formulation on<br>PSA response | Percent change in PSA from baseline (prior to injection) at Week 12 and Week 24 (Percent change in PSA is defined as the absolute value of difference between the PSA values at Week 12 and Week 24 and the baseline value divided by the baseline value) |
| To assess the PK of triptorelin pamoate 22.5 mg 6-month formulation in a subset of 12 participants | PK parameters for dosing interval up to 24 weeks: t <sub>max</sub> , C <sub>max</sub> , AUC <sub>0-169</sub> AUC <sub>last</sub> |
| To assess the PD of testosterone in a subset of 12 participants | PD parameters for dosing interval up to 24 weeks: t <sub>max</sub> , C <sub>max</sub> t <sub>cast</sub> |
| To assess the PK of triptorelin pamoate 22.5 mg 6-month formulation for all participants | <ul> <li>Sparse plasma concentrations of triptorelin<br/>at pre-dose and at Week 4, 8, 12, 16, 20 and<br/>24</li> </ul> |
| To assess the PD of testosterone for all participants | Sparse serum concentrations of testosterone<br>at pre-dose and at Week 4, 8, 12, 16, 20 and<br>24 |
| Exploratory | |
| To evaluate the PK/PD relationship between<br>the PK of triptorelin pamoate 22.5 mg<br>6-month and testosterone concentration<br>versus time profiles (PD) | o the visit on Day 169: AUC₁₅₅≔area under the plasma concentration time |

AUC<sub>0-169</sub>=area under the plasma concentration time curve from time 0 to the visit on Day 169; AUC<sub>last</sub>=area under the plasma concentration time curve from time 0 to the last quantifiable concentration; C<sub>max</sub>=maximum concentration; ECG=electrocardiogram; PD=pharmacodynamics; PK=pharmacokinetics; PSA=prostate specific antigen; t<sub>cast</sub>=time to castration; TEAE=treatment-emergent adverse event; t<sub>max</sub>=time to peak serum/plasma concentration

Note:  $\hat{A}$  list of laboratory parameters to be assessed during the study are presented in Appendix 10.2.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 18/92

#### **Overall Design:**

This is a prospective, interventional, multicentre, open-label phase IIIb, single-arm study with a treatment period of 24 weeks for each participant. A total of 195 Chinese adult participants with locally advanced or metastatic prostate cancer will be enrolled in the study. All enrolled participants will receive one intramuscular (i.m.) injection of the 6-month formulation containing 22.5 mg triptorelin pamoate on Day 1.

#### **Intervention Groups and Duration:**

Triptorelin pamoate 22.5 mg (6-month formulation), i.m. injection, single dose on Day 1.

#### **Visit Frequency:**

This study will consist of a 4-week screening period, a single open-label administration of the study intervention on Day 1. Following treatment, visits will occur on Day 2, Day 3, Day 5, Day 8, Day 15, Day 22 in a subset of 12 participants, and for all participants on Day 29, Day 57, Day 85, Day 113, Day 141 and Day 169.

### **Study Participant Duration:**

Participants are expected to participate in this study for 24 weeks.

#### **Number of Participants:**

Approximately 195 participants (including a rich sampling pharmacokinetic/pharmacodynamic subset of 12 participants) are planned to be assigned to study intervention.

#### **Statistical Methods:**

Sample Size Determination

The sample size was estimated based on data from the previous Study DEB-TRI6M-301, 97.5% of participants achieving castration on Day 29 and 93% of participants maintaining castration from Week 8 to Week 24.

Sample size is calculated to fulfil the co-primary efficacy criteria of this study, which is to assess the proportion of participants achieving castrate levels of testosterone on Day 29 and the proportion of participants maintaining the castrate levels of serum testosterone from Week 8 to end of Week 24.

For an exact binomial test of a proportion with a two-sided nominal significance level of 0.05 and null proportion of 85%, a sample size of 165 participants has an exact power of 88.3% when the true proportion is 93% (of participants maintaining castration from Week 8 to Week 24). This sample size of 165 participants has a power >99.9% when the true proportion is 97.5% (of participants achieving castrate testosterone levels). Exact two-sided 95% CI for a binomial proportion was computed by statistical analysis software (SAS) using the exact binomial distributions.

Assuming the dropout rate will be around 15%, a sample size of 195 participants with locally advanced or metastatic prostate cancer in total is planned for this study.

#### Primary Analysis

The analysis sets for the primary and secondary efficacy endpoints will be the full analysis set (FAS) and the per protocol (PP) set.

Co-primary endpoints will be tabulated with two-sided 95% confidence interval (95% CI) using the Clopper-Pearson exact method.

#### Secondary Analyses

Prostate-specific antigen (PSA) percent change from pre-treatment Day 1 will be reported at Week 12 and Week 24, using descriptive statistics. The PK (triptorelin) and PD (testosterone) metrics will be reported as descriptive statistics.

For the analysis of safety, any participant who receives the single dose of triptorelin will be analysed (Safety population). The incidence of AEs as per National Cancer Institute – Common Toxicity Criteria (NCI-CTCAE) Version 5.0 grading will be summarised by System Organ Class (SOC), preferred term (PT) severity and relationship to study drug. Adverse events will be coded using Medical Dictionary of Drug Regulatory Activities (MedDRA) Version 24.1 (or higher if available) prior to analysis. Changes from baseline in clinical laboratory tests, physical examinations, electrocardiogram (ECG) and vital signs will be summarised using descriptive statistics.

The data will be summarised with the descriptive statistics (i.e. N, means, standard deviation, minimum, maximum, median) for the continuous variables and with counts and percentages for the categorical variables. In addition, for PK endpoints, the geometric mean, the standard deviation of the geometric mean, and geometric coefficient of variance% will be presented.

#### 1.2 Schema

The study schema is shown in Figure 1.

#### Figure 1 Study Schema



PD=pharmacodynamic; PK=pharmacokinetic; Q4W=every 4 weeks

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 **PAGE 20/92** 

#### **Schedule of Activities (SoA)** 1.3

The schedule of activities during the study is summarised for all participants in Table 1, except the PK/PD subset of 12 participants which is summarised in Table 2.

If the Coronavirus Disease 2019 (COVID-19) pandemic prevents participants from coming to the site, participants can have their study visit assessments performed remotely as judged appropriate by the investigator. This must be discussed with the sponsor before being implemented. In such a case, the investigator will perform a telemedicine visit and will make every effort, where applicable, to contact the participant's general practitioner or specialist physician to ensure all important medical information and safety event(s) occurring since the last visit are collected. Guidance on how to collect protocol-planned assessments will be provided to the investigator in a separate document. Such document will be filed in the trial master file. Independent ethics committees (IECs)/institutional review boards (IRBs) will be notified of the changes as applicable locally. Of note, as the adapted visit deviates from the regular protocol plan, the changes will be recorded as protocol deviations related to COVID-19.

Table 1 Schedule of Activities for All Participants Except the Pharmacokinetic/Pharmacodynamic Subset

| Procedure | Screening | | | Intervent | tion Period | | | EoS/EW |
|---|---|---|---|---|---|---|---|---|
| End of Week | - | - | Week 4 | Week 8 | Week 12 | Week 16 | Week 20 | Week 24 |
| Day | D-28 to D-1 | D1 | D29 | D57 | D85 | D113 | D141 | D169 |
| Visit Window | - | - | ±3 days | ±3 days | ±3 days | ±3 days | ±3 days | ±3 days |
| Informed consent | X | | | | | | | |
| Eligibility | X | X | | | | | | |
| Demography | X | | | | | | | |
| Medical and surgical history | X | | | | | | | |
| Physical examination [f] | X | X [a] | | | X | | | X |
| MRI scan [g] | X | | | | | | | |
| Disease-specific medical history | X | | | | | | | |
| Prior disease-specific treatment | X | | | | | | | |
| Body weight | X | | | | | | | X |
| Vital signs | X | X [a] | X | X | X | X | X | X |
| 12-lead electrocardiogram[b] | X | | X | | | | | X |
| ECOG Score | X | | | | | | | |
| Injection triptorelin 6M | | X | | | | | | |
| Blood samples for triptorelin PK | | X [a] | X | X | X | X | X | X |
| Blood sample for testosterone PD [h] | X | X [a, e] | X | X | X | X | X | X |
| Blood samples for PSA [h] | X | X [a, e] | | | X | | | X |
| Blood samples [c] laboratory safety tests | X | X [a, e] | | | | | | X |
| Local tolerance [d] | | X | | | | | | |
| Previous (excluding disease-specific) and concomitant medication | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X |

6M=6-month formulation, AE=adverse event, ALT=alanine aminotransaminase, AST=aspartate aminotransaminase, CRF=case report form, D=day; ECG=electrocardiography; ECOG=Eastern Cooperative Oncology Group, EoS/EW=end of study/early withdrawal, Hb=haemoglobin, M1b=distant metastasis bone(s), MRI=magnetic resonance imaging; PD=pharmacodynamic, PK=pharmacokinetics, PSA=prostate-specific antigen, WBC=white blood cell.

#### PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024


- a Assessment or blood sampling to be performed prior to study intervention injection. PK Predose sampling window ( $\leq$ 30 minutes).
- b ECG to be assessed as clinically indicated at any other time in the study as required.
- c Haematology (WBC, platelet count, Hb), Blood Chemistry (creatinine, glucose, ALT, AST, alkaline phosphatase, bilirubin (total and conjugated)) will be tested at the local laboratory. Glucose: fasting levels in all participants at Screening visit, fasting levels on Days 1 and 169. Fasting is not necessary for diabetic participants.
- d Injection site to be specifically checked 2 hours ±15 minutes after injection for local reactions on Day 1. After Day 1, any local reaction AE to be collected on the CRF in the same manner as other AEs.
- e Measurement of testosterone, PSA and laboratory safety tests for analysis purposes only and not for eligibility. The screening testosterone, PSA and safety laboratory test results will be used for eligibility.
- f Complete physical examination to be performed (or brief physical examination based on investigator judgement). Participants, particularly those with M1b status, should be advised regarding clinical signs suggestive of spinal cord compression.
- g Scan for prostate gland or the whole body, only if necessary, based on investigator's judgement. An MRI scan is not required if performed within 1 month of screening.
- h Testosterone and PSA testing will be performed at the central laboratory.

See Appendix 10.5 for ECOG performance scale.

 Table 2
 Schedule of Assessments for the Pharmacokinetic/Pharmacodynamic Subset of Participants

| Procedures | Screening | | | | | In | tervent | tion Pe | riod | | | | | EoS/EW |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| End of Week | - | - | - | - | - | - | - | - | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>24 |
| Day | D-28 to<br>D-1 | D1 | D2 | D3 | D5 | D8 | D15 | D22 | D29 | D57 | D85 | D113 | D141 | D169 |
| Visit Window | | | | | | | | | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days |
| Informed consent | X | | | | | | | | | | | | | - |
| Eligibility | X | X | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | |
| Medical and surgical history | X | | | | | | | | | | | | | |
| Physical examination [g] | X | X [a] | | | | | | | | | X | | | X |
| MRI scan [h] | X | | | | | | | | | | | | | |
| Disease-specific medical history | X | | | | | | | | | | | | | |
| Prior disease-specific treatment | X | | | | | | | | | | | | | |
| Body weight | X | | | | | | | | | | | | | X |
| Vital signs | X | X [a] | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-lead electrocardiogram[b] | X | | | | | | | | X | | | | | X |
| ECOG Score | X | | | | | | | | | | | | | |
| Injection triptorelin 6M | | X | | | | | | | | | | | | |
| Blood sample for triptorelin PK | | X [c] | X | X | X | X | X | X | X | X | X | X | X | X |
| Blood sample for testosterone PD [i] | X | X [a, f] | X | X | X | X | X | X | X | X | X | X | X | X |
| Blood sample for PSA [i] | X | X [a, f] | | | | | | | | | X | | | X |
| Blood samples for [d] laboratory safety tests | X | X [a, f] | | | | | | | | | | | | X |
| Local tolerance [e] | | X | | | | | | | | | | | | |


#### PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024

| Procedures | Screening | | | | | Int | tervent | ion Pe | riod | | | | | EoS/EW |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| End of Week | - | - | - | - | - | - | - | - | Week<br>4 | Week<br>8 | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>24 |
| Day | D-28 to<br>D-1 | D1 | D2 | D3 | D5 | D8 | D15 | D22 | D29 | D57 | D85 | D113 | D141 | D169 |
| Visit Window | | | | | | | | | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days | ±3<br>days |
| Previous (excluding disease-specific) and concomitant medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

6M=6-month formulation, AE=adverse event, ALT=alanine aminotransaminase, AST=aspartate aminotransaminase, CRF=case report form, D=day; ECG=electrocardiography; ECGG=Eastern Cooperative Oncology Group, EoS/EW=end of study/early withdrawal; h=hours; Hb=haemoglobin, M1b=distant metastasis bone(s); MRI=magnetic resonance imaging; PD=pharmacodynamic, PK=pharmacokinetics, PSA=prostate-specific antigen, WBC=white blood cell.

- a Assessment or blood sampling to be performed prior to study intervention injection.
- b ECG to be assessed as clinically indicated at any other time in the study as required.
  - Sampling on Day 1. PK time sampling windows:
    - Pre-dose (\le 30 mins) prior to study drug injection
    - 1h, 2h, 3h post-dose  $\pm 5$  mins
    - 4h, 6h, 8h post-dose  $\pm 15$  mins
    - 12h post-dose  $\pm 30$  mins
    - 24h post-dose  $\pm 1$  hour
    - 48h post-dose  $\pm 2$  hours
    - 96h post-dose ±3 hours
    - 168h post-dose ±4 hours
    - Day 15 (2 weeks post-dose)  $\pm 24$  hours
    - Day 22 (3 weeks post-dose)  $\pm 24$  hours
    - Day 29, 57, 85, 113, 141, 169 = clinic visit time windows ( $\pm 3$  days)
- d Haematology (WBC, platelet count, Hb), Blood Chemistry (creatinine, glucose, ALT, AST, alkaline phosphatase, bilirubin (total and conjugated) will be tested at the local laboratory. Glucose: Fasting levels in all participants at Screening visit, fasting levels on Days 1 and 169. Fasting is not necessary for diabetic participants.
- e Injection site to be specifically checked 2 hours ±15 minutes after injection for local reactions on Day 1. After Day 1 any local reaction AEs to be collected on the CRF in the same manner as other AEs.
- f Measurement of testosterone, PSA and laboratory safety tests for analysis purposes only and not for eligibility. The screening testosterone, PSA and safety laboratory test results will be used for eligibility.
- g Complete physical examination to be performed (or brief physical examination based on investigator judgement). Participants, particularly those with M1b status, should be advised regarding clinical signs suggestive of spinal cord compression.
- h Scan for prostate gland or the whole body, only if necessary, based on investigator's judgement. An MRI scan is not required if performed within 1 month of screening.
- i Testosterone and PSA testing will be performed at the central laboratory.

See Appendix 10.5 for ECOG performance scale.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 25/92

#### 2 INTRODUCTION

Triptorelin is an agonist analogue of natural GnRH. The principal modification consists of substitution of natural glycine in position 6 by a D-amino acid (D tryptophan). Clinical and animal studies have provided positive results of triptorelin's action in hormone-dependent disorders such as prostate cancer, endometriosis, central precocious puberty, uterine fibromyomas, in vitro fertilisation and breast cancer.

# 2.1 Study Rationale

Results from a global phase III study have shown that the new triptorelin 6-month formulation (22.5 mg) was well tolerated and rapidly induced and maintained castration in participants with locally advanced or metastatic prostate cancer [Lundstrom 2009].

The advantage of the sustained-release 6-month triptorelin pamoate formulation is that the reduced frequency of injections will provide greater convenience to both the patient and the physician and may also improve patient acceptability and compliance with the injection schedule.

The present study will assess the efficacy and safety of the sustained-release 6-month triptorelin pamoate formulation in Chinese participants with locally advanced or metastatic prostate cancer for confirming the registration of this product in China. In addition, triptorelin pharmacokinetics (PK) and testosterone pharmacodynamics (PD) will be assessed in the study population.

# 2.2 Background

Prostate cancer is one of the most commonly occurring malignancies in the male population and thus the second cause of death from cancer in men over 50 in the western world. In most patients, it is an androgen-dependent tumour at initial presentation.

Growth of the prostatic tissue is regulated by a network of hormones in which androgens play a major role. Gonadotropin-releasing hormone (GnRH), also known as luteinizing hormone releasing hormone (LHRH), released in a pulsatile manner by the hypothalamus, stimulates the pituitary to release in pulses the gonadotropins luteinizing hormone (LH) and follicle stimulating hormone (FSH). LH stimulates the production of testicular testosterone; however, approximately 5% of circulating testosterone is independently produced by the adrenal glands. FSH plays a role in the regulation of spermatogenesis.

Since the pioneering studies of Huggins and Hodges [1941, 1941a] in the 1940's about the regulatory role played by the testicular androgens in the growth of prostate cancer cells, the mainstay of treatment for advanced prostate cancer was for decades androgen deprivation by bilateral orchiectomy and/or oestrogen therapy. The limitations of these therapeutic modalities led to the development of GnRH agonists, which have made medical castration the preferred option among many patients with metastatic disease [Filicori 1994]. The efficacy and safety of these agents is now well established, and GnRH agonists are not associated with an increased risk of cardiovascular disease.

The therapeutic activity of the GnRH agonists is through pituitary down-regulation of their own receptors achieved by continuous and chronic administration, providing almost complete suppression of LH and FSH secretion leading to suppression of testicular function.

Achievement of castration levels of testosterone is generally obtained around one month after start of therapy. Of note, long term endocrine status and evolution of advanced prostate cancer treated with GnRH agonists are similar to those observed after surgical castration [Parmar 1987, DeSy 1988, Botto 1987] but in contrast to surgical castration, treatment with GnRH agonists initially results in a markedly, albeit temporary (~2 weeks), increase of gonadal androgen

release (flare-up phenomenon). The initial rise in testosterone may cause a temporary worsening of symptoms including increase in bone pain within the first days of treatment; for these reasons, GnRH agonists are contraindicated for use in patients presenting metastases with neurologic symptomatology, or other possible life-threatening metastases. The most significant side effects - hot flushes, decreased libido and erectile dysfunction - are linked to the pharmacological effect (castrate levels of testosterone) and are usually relatively mild and reversible upon cessation of therapy.

Since the discovery and synthesis of GnRH, many analogues of the native decapeptide have been synthesised in attempts to develop agonists with increased in vivo half-life and potency.

As shown in the amino acid sequences below, the major structural difference between the native decapeptide and the triptorelin agonist is the substitution of a different D-amino acid at position six, which is the hinge between the two active portions of the peptide. However, triptorelin retains the parts of the native decapeptide responsible for its biological activity.

Decapeptide

10 Glu-His-Trp-Ser-Tyr- Gly -Leu-Arg-Pro-Gly-NH2

Triptorelin

(pyro) Glu-His-Trp-Ser-Tyr- D-Trp -Leu-Arg-Pro-Gly-NH2

GnRH has a L-glycine at position six, whereas triptorelin has a D-tryptophan. The substitution of the D-amino acid increases resistance to cleavage by proteolytic enzymes and increases biological potency relative to the native decapeptide [Barron 1982]. Triptorelin, like other GnRH agonists, has a short half-life in vivo (t½=5 h), therefore, sustained-release dosage forms have been developed by combining the peptide with a biocompatible and biodegradable copolymer (lactide-glycolide). By modifying the molar ratio of lactic acid to glycolic acid, the peptide is released continuously over periods ranging from 28 days (1-month formulation) to 168 days (6-month formulation) following administration of a single intramuscular (i.m.) injection.

The 6-month triptorelin formulation (22.5 mg) has been evaluated in a multicentre, non-comparative phase III study in participants with advanced prostate cancer, conducted between July 2006 and August 2007 [Lundstrom 2009]. The results from the study have shown that the new triptorelin 6-month formulation (22.5 mg) rapidly induces and maintains castration in participants with locally advanced or metastatic prostate cancer. In the intention-to-treat (ITT) population, 97.5% (117/120) of participants were castrated (testosterone level <50 ng/dL) on Day 29, and 93.0% (107/115) of participants maintained castration from Week 8 (Day 57) to end of Week 48. The efficacy results of the 6-month formulation have been reviewed with those obtained in previous studies with the marketed triptorelin 1- and 3-month formulations. Results show that the rate of castration achieved with the 6-month formulation on Day 29, after the first triptorelin injection, was comparable to those with the 1-month and 3-month formulations [Breul 2017].

In terms of local tolerance at the injection site, intramuscular triptorelin injections were well tolerated and in the phase III study where injection site reactions were assessed by active questioning: 6.7% participants with injection-site reactions reported as adverse events (AEs), which is lower than for other 6-month GnRH formulations [Lundstrom 2009]. In a pooled analysis, very few (<5%) local adverse reactions at the injection site have been reported in clinical studies with all triptorelin sustained-release formulations (1-, 3- and 6-month) [Breul 2017].

A more detailed description of the product, including further details on administration procedures and dosage are provided in Section 6.

#### 2.3 Benefit/Risk Assessment

Detailed information about the known and expected benefits and risks and reasonably expected AEs of triptorelin may be found in the IB.

#### 2.3.1 Risk Assessment

A risk assessment for this study is provided in Table 3.

Table 3 Study Risk Assessment

| Potential Risk of Clinical<br>Significance | Summary of Data/Rationale for<br>Risk | Mitigation Strategy |
|---|---|---|
| Study Intervention: Triptorelin | | |
| There is no major known nonclinical risk associated with the study intervention Clinical risks associated with the study intervention in may include: • hot flushes • erectile dysfunction • loss of libido • impaired physical activities • metabolic syndrome • cardiovascular events • anxiety/depression • decreased bone mineral density • risk of abortion or foetal abnormality [a] See Section 8.3 | See IB Section 6.6.1 | Participant selection: Participants with significant medical conditions and at high risk of presenting treatment related SAEs and high-grade toxicity will be excluded from the study. Participant monitoring: During the study, there will be close monitoring of the participants for safety including local tolerability (see Section 8.3.6) Withdrawal criteria: Participants who become at risk of unacceptable toxicity will be withdrawn from the study intervention. |
| | Study Procedures | |
| There are no specific risks related to the study design or procedures. | All procedures requested for the study are commonly used in clinical practice and the design does not create any specific risk or delay possible therapeutic option for participants | Not applicable |

IB=investigator's brochure; SAE=serious adverse event

# 2.3.2 Benefit Assessment

Based on the nonclinical and clinical data generated up to finalisation of the protocol, treatment with triptorelin 6-month formulation may maintain castrate levels of testosterone for a longer period, i.e. 6 months (24 weeks), thereby reducing the need for frequent injections, in Chinese participants with locally advanced or metastatic prostate cancer to a similar extent as in a previous global phase III study.

a Pregnancy is not relevant in this study population. However, reproductive risks are listed for completeness for female partners of participants who may become pregnant.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 28/92

### 2.3.3 Overall Benefit: Risk Conclusion

Taking into account the measures taken to minimise risk to participants, the potential risks identified in association with triptorelin are justified by the anticipated benefits that may be afforded to Chinese participants with locally advanced or metastatic prostate cancer.

### 3 OBJECTIVES AND ENDPOINTS

Table 4 Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the efficacy of triptorelin pamoate 22.5 mg 6-month formulation in achieving castrate levels of testosterone To evaluate the efficacy of triptorelin pamoate 22.5 mg 6-month formulation in maintaining the castrate levels of serum | <ul> <li>Percentage of participants achieving castrate levels of serum testosterone (&lt;50 ng/dL or 1.735 nmol/L) on Day 29</li> <li>Percentage of participants maintaining the castrate levels from Week 8 to Week 24</li> </ul> |
| testosterone | |
| To assess the safety profile including local tolerability of triptorelin pamoate 22.5 mg 6-month formulation | <ul> <li>Incidence of TEAEs (including local tolerability) throughout the study i.e., up to Week 24</li> <li>Change from baseline in clinical safety laboratory parameters (blood chemistry and haematology) at Week 24</li> <li>Change from baseline in physical examination at Day 1, Week 12 and Week 24</li> <li>Change from baseline in ECG at Week 4 and Week 24</li> <li>Change from baseline in vital signs (blood pressure and heart rate) at each visit up to Week 24</li> </ul> |
| To demonstrate the effect of triptorelin<br>pamoate 22.5 mg 6-month formulation on<br>PSA response | Percent change in PSA from baseline (prior to injection) at Week 12 and Week 24 (percent change in PSA is defined as the absolute value of difference between the PSA values at Week 12 and Week 24 and the baseline value divided by the baseline value) |
| To assess the PK of triptorelin pamoate 22.5 mg 6-month formulation in a subset of 12 participants | PK parameters for dosing interval up to 24 weeks: t <sub>max</sub> C <sub>max</sub> AUC <sub>0-169</sub> AUC <sub>last</sub> |
| To assess the PD of testosterone in a subset of 12 participants | <ul> <li>PD parameters for dosing interval up to 24 weeks: <ul> <li>t<sub>max</sub></li> <li>C<sub>max</sub></li> <li>t<sub>cast</sub></li> </ul> </li> </ul> |
| To assess the PK of triptorelin pamoate 22.5 mg 6-month formulation for all participants | <ul> <li>Sparse plasma concentrations of triptorelin<br/>at pre-dose and post-dose at Weeks 4, 8, 12,<br/>16, 20 and 24</li> </ul> |
| To assess the PD of testosterone for all participants | <ul> <li>Sparse serum concentrations of testosterone<br/>at pre-dose and post-dose at Weeks 4, 8, 12,<br/>16, 20 and 24</li> </ul> |
| Exploratory | |
| To evaluate the PK/PD relationship between<br>the PK of triptorelin pamoate 22.5 mg<br>6-month formulation and testosterone<br>concentration versus time profiles (PD) | m time 0 to the visit on Day 169: AUClast=area under the |

AUC<sub>0-169</sub>=area under the plasma concentration time curve from time 0 to the visit on Day 169; AUC<sub>last</sub>=area under the plasma concentration time curve from time 0 to the last quantifiable concentration; C<sub>max</sub>=maximum concentration;

IPSEN GROUP D-CN-52014-237

# CONFIDENTIAL PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024


ECG=electrocardiogram; PD=pharmacodynamics; PK=pharmacokinetics; PSA=prostate specific antigen;  $t_{cast}$ =time to castration; TEAE=treatment-emergent adverse event;  $t_{max}$ =time to peak serum/plasma concentration Note: A list of laboratory parameters to be assessed during the study are presented in Appendix 10.2.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 31/92

#### 4 STUDY DESIGN

#### 4.1 Overall Design

This is a prospective, interventional, multicentre, open-label phase IIIb, single-arm study with a treatment period of 24 weeks for each participant. A total of 195 Chinese adult participants with locally advanced or metastatic prostate cancer will be enrolled in the study. All enrolled participants will receive one i.m. injection of the 6-month formulation containing 22.5 mg triptorelin pamoate on Day 1.

This study will consist of a 4-week screening period, during which participants with advanced or metastatic prostate cancer will be screened for eligibility. On Day 1, eligible participants will receive a single open-label administration of the study intervention. Following treatment on Day 1, visits will occur on Day 2, Day 3, Day 5, Day 8, Day 15, Day 22 in a subset of 12 participants, and for all participants on Day 29, Day 57, Day 85, Day 113, Day 141 and Day 169. For more details on sampling schedule see the SoA (Table 1 and Table 2).

The maximum duration of the study is approximately 30 months from screening to the last study visit. Participants who complete all scheduled visits will be considered to have completed the study. Participants who complete the study will have final procedures and assessments performed at the final visit (Day 169). Participants who withdraw from the study before the completion of the Day 169 evaluation period will have early discontinuation procedures and assessments performed at their final visit.

The study design is illustrated in Figure 1.

# 4.2 Scientific Rationale for Study Design

This single-arm, phase III study will investigate the efficacy, safety and PK/PD of triptorelin 6-month formulation in Chinese adult males with locally advanced or metastatic prostate cancer.

According to data from China National Cancer Registration Institute, prostate cancer has become the most common tumour in male urinary malignancies since 2008. The incidence rate was approximately 9.80/100,000 in 2014 and ranks the sixth common malignancy in male malignant tumours. The mortality of prostate cancer is 4.22/100,000, and it is the 9th common cause of death in all male malignancies. The staging varies widely between China and Western developed countries. In China, only 30% of newly diagnosed patients are clinically localised, and the rest are locally advanced or extensively metastatic disease, who have lost the chance of radical treatment with poor prognosis [National Health Commission China 2019]. This study will enrol adult Chinese men with advanced prostate cancer.

The non-comparative, open-label clinical study design is acceptable as the efficacy of triptorelin will be assessed by the percentage of participants achieving castrate levels of serum testosterone (defined as <50 ng/dL or 1.735 nmol/L) on Day 29 and maintaining castrate levels of serum testosterone from Week 8 to Week 24 (co-primary endpoints). Studies conducted in Western countries have shown that the rate of castration achieved with the 6-month formulation on Day 29, after the first triptorelin injection, was comparable to those with the 1-month and 3-month formulations [Breul 2017]. No studies have evaluated the 6-month triptorelin formulation in Chinese men with locally advanced or metastatic prostate cancer, thus the outcomes of this study intend to fulfil an unmet need and provide treatment convivence for the patient and physician.

This study will evaluate the PK/PD profile of triptorelin 6-month formulation in this study population. The blood sample collection scheme was designed to collect the minimum number of blood samples to help provide useful PK/PD information of study treatment in Chinese men with locally advanced or metastatic prostate cancer.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 32/92

#### 4.3 **Justification for Dose**

For this intervention, the term "dose" refers to the i.m. injection of triptorelin 22.5 mg created to guarantee the release of a monthly dose of 3.75 mg over a 169-day period. In addition, results from a phase III study have shown the 6-month triptorelin 22.5 mg formulation to induce and maintain castration in participants with locally advanced or metastatic prostate cancer, as well as demonstrate a good safety profile [Lundstrom 2009].

### 4.4 End of Study Definition

The end of the study (EoS) is defined as the date of the last visit of the last participant in the study as shown in the SoA (Table 1 and Table 2).

The overall duration of the study (from first participant in, to last participant out) will be approximately 30 months. The study will be considered to have ended after the last participant has completed the last visit (at Week 24) in the study.

A participant is considered to have completed the study if they have completed all phases of the study including the last visit.

Criteria for study intervention discontinuation and participant discontinuation/withdrawal from the study are described in Section 7.1 and Section 7.2, respectively. Loss to follow-up is described in Section 7.3.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 33/92

#### 5 STUDY POPULATION

Prospective approval of protocol deviations to recruitment and enrolment criteria, also known as protocol waivers or exemptions, is not permitted.

#### 5.1 Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

- 1. Participant is capable of giving signed informed consent as described in Appendix 10.1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
- 2. Participant must be over 18 years of age, at the time of signing the informed consent.
- 3. Has a histologically or cytologically confirmed adenocarcinoma, locally advanced or metastatic prostate cancer, which is staged T<sub>3-4</sub>N<sub>x</sub>M<sub>0</sub> or T<sub>x</sub>N<sub>1</sub>M<sub>0</sub> or T<sub>x</sub>N<sub>x</sub>M<sub>1</sub> according to the TNM classification (Appendix 10.4). Or participant has PSA recurrence after curative treatment and be a candidate for androgen deprivation therapy (ADT).
  - (Note: PSA recurrence after radical prostatectomy: PSA ≥0.2 ng/mL and rising, confirmed on a repeat test; PSA recurrence after radiation therapy: PSA increased 2 ng/mL than the lowest level.)
- 4. Has serum testosterone level >150 ng/dL (> 5.2 nmol/L).
- 5. Has expected survival time  $\geq$ 12 months according to the investigator's assessment.
- 6. Has Eastern Cooperative Oncology Group (ECOG) performance status score ≤1 (see Appendix 10.5).
- 7. Has absence of another malignancy, other than local dermatological, for the previous 5 years.
- 8. Participant is male.
- 9. Male participants must agree that, if their partner is at risk of becoming pregnant, they will use an effective method of contraception. The participant must agree to use the contraception during the whole period of the study and for 9 months after the last dose of study intervention.

#### 5.2 Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

Medical conditions

- 1. Risk of a serious complication in the case of tumour flare (known or suspicion of vertebral metastases threatening spinal cord compression or significant obstructive uropathy).
- 2. Presence of another neoplastic lesion or brain metastases.
- 3a. Previous history of QT prolongation or concomitant use of medicinal products known to prolong the QT interval or with a known risk of torsades de pointes.
- 4a. Metastatic hormone-sensitive prostate cancer with high tumour burden. (Note: high tumour burden: presence of visceral metastases and/or at least four bone lesions with at least one lesion outside the vertebral column and/or pelvis per CHAARTED study (Kyriakopoulos 2018).
- 5. Metastatic castration-resistant prostate cancer.

#### Prior/concomitant therapy

6. Previous surgical castration.

- 7a. Previous hormone therapy (including abiraterone) for prostate cancer within 6 months prior to study screening.
- 8a. Previous cytotoxic chemotherapy treatment within 6 months prior to study screening.
- 9a. Use of finasteride or dutasteride within 2 months prior to study screening.
- 10. Previous hypophysectomy or adrenalectomy.
- 11a. Any current use or use within 6 months prior to treatment start of medications which are known to affect the metabolism and/or secretion of androgenic hormones: ketoconazole, aminoglutethimide, oestrogens and antiandrogens.
  - Note: antiandrogen: enzalutamide, apalutamide or darolutamide is allowed (if required per investigator's clinical judgement) due to no interference on the metabolism and/or secretion of androgenic hormones.
- 12a. Current use of systemic or inhaled corticosteroids (topical application permitted).
- 13. Any previous use of traditional Chinese medicine or herbal products within 1 month prior to study screening or planned use during the study of products, which are known to have cytotoxic effect or affect the metabolism and/or secretion of androgenic hormones.

#### Prior/concurrent clinical study experience

14a. Participation in another study with an investigational drug or treatment within 3 months prior to study screening or within 5 drug half-lives of the investigational drug (whichever is the longer).

# Diagnostic assessments

15. Severe kidney or liver impairment (creatinine >2 x upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >3 x ULN).

#### Other exclusions

- 16. Any concomitant disorder or resulting therapy that is likely to interfere with participant compliance, the i.m. administration of the drug or with the study in the opinion of the investigator.
- 17. Known hypersensitivity to triptorelin or any of its excipients, GnRH, other GnRH agonist/analogues.
- 18. Known active use of recreational drug or alcohol dependence in the opinion of the investigator.

#### 5.3 **Lifestyle Considerations**

Participants will be advised to avoid chronic alcohol use and smoking during the study.

#### 5.4 **Screen Failures**

A screen failure occurs when a participant who consents to participate in the clinical study is not subsequently entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes date of informed consent, demography, reason for screen failure, eligibility criteria and any serious adverse event (SAE).

Individuals who do not meet the criteria for participation in this study (screen failure) will not be rescreened.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 35/92

#### 6 STUDY INTERVENTION AND CONCOMITANT THERAPY

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

#### 6.1 Study Intervention(s) Administered

Study intervention is described in Table 5.

Table 5 Study intervention administered

| Intervention Name | Triptorelin pamoate (embonate) salt |
|---|---|
| <b>Intervention Description</b> | A PR formulation of triptorelin pamoate 6-month formulation in D,L-lactide-co-glycolide polymers for single i.m injection |
| Type | Drug |
| Dose Formulation | A yellow freeze-dried cake or powder supplied in a single 6 mL glass vial |
| Unit Dose Strength(s) | 22.5 mg (with release of a monthly dose of 3.75 mg over a 169-day period) |
| Dosage Level(s) | Single dose delivered on Day 1 |
| Route of Administration | i.m. injection |
| Use | Experimental |
| IMP and NIMP/AxMP | IMP |
| Sourcing | Manufactured by Debiopharm and provided centrally by the sponsor |
| Packaging and Labelling | Study intervention will be provided in a box containing one vial, one ampoule and one blister containing one injection syringe and two injection needles. Each box will be labelled as required per country requirement. |
| Storage requirements | To be stored in the outer carton at a temperature below 25°C in a dry place, protected from freezing |
| Current Name | Diphereline® |

i.m.=intramuscular; IMP=investigational medicinal product; NIMP=non-investigational medicinal product; AxMP=auxiliary medicinal product; PR=prolonged release

### 6.2 Preparation, Handling, Storage and Accountability

The investigator or an approved representative (e.g. pharmacist) will ensure that triptorelin is reconstituted and dispensed by a member of staff specifically authorised by the Investigator and trained for the IMP reconstitution and administration.

The suspension for injection must be reconstituted using an aseptic technique and only using the ampoule of solvent for injection.

The instructions for reconstitution hereafter and in the leaflet provided with triptorelin must be strictly followed.

The solvent should be drawn into the syringe provided using the reconstitution needle (20 G, without safety device) and transferred to the vial containing the powder. The suspension should be reconstituted by swirling the vial gently from side to side for long enough until a homogeneous, milky suspension is formed. Do not invert the vial.

It is important to check there is no unsuspended powder in the vial. The suspension obtained should then be drawn back into the syringe, without inverting the vial. The reconstitution needle should then be changed, and the injection needle (20 G, without safety device) used to administer the product.

As the product is a suspension, the injection should be administered for a single use <u>immediately</u> after reconstitution to prevent precipitation.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 36/92

- The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study intervention received and any discrepancies are reported and resolved before use of the study intervention.
- Only participants screened in the study and who meet the eligibility criteria may receive study intervention and only authorised site staff may supply or administer study intervention. All study intervention must be stored in a secure, environmentally controlled and monitored (manual or automated) area in accordance with the labelled storage conditions with access limited to the investigator and authorised site staff.
- The investigator, institution or the head of the medical institution (where applicable) is responsible for study intervention accountability, reconciliation, and record maintenance (i.e. receipt, reconciliation and final disposition records).
- The sponsor will provide guidance on the destruction of unused study intervention. If destruction is authorised to take place at the investigational site, the investigator must ensure that the materials are destroyed in compliance with applicable environmental regulations, institutional policy and any special instructions provided by the sponsor. All destruction must be adequately documented.

Further guidance and information for the receipt, preparation, management and disposal/return of the study intervention are provided in the "Investigational Medicinal Product Handling Manual".

### 6.3 Measures to Minimize Bias: Randomisation and Blinding

#### 6.3.1 Randomisation

This is a non-randomised, open-label study.

#### 6.3.2 Maintenance of Blinding

This is an open-label study therefore no procedures for blinding are applicable.

#### 6.4 Study Intervention Compliance

When participants are dosed at the site, they will receive study intervention directly from the investigator or designee, under medical supervision. The date and time of each dose administered in the site will be recorded in the source documents and in the electronic case report form (eCRF). The dose of study intervention and study participant identification will be confirmed at the time of dosing by a member of the study site staff other than the person administering the study intervention.

#### **6.5** Dose Modification

Not applicable. No dose modifications are to be performed in the study.

### 6.6 Continued Access to Study Intervention after the End of the Study

The participants will not receive any additional study intervention following the end of the study.

#### **6.7** Treatment of Overdose

The pharmaceutical properties of triptorelin 6-month formulation and its mode of administration make accidental or intentional overdose unlikely. There is no experience of overdose from clinical studies (for more information see the summary of product characteristics). If overdose occurs, this should be managed symptomatically.

In the event of an overdose, the investigator should:

• Contact the medical monitor immediately.
- Closely monitor the participant for any AE/SAE and laboratory abnormalities (at least up to the Week 24 visit).
- Document the quantity of the excess dose as well as the duration of the overdose. See Section 10.3.1 for reporting requirements concerning overdose.

#### 6.8 **Concomitant Therapy**

Any medication (excluding prior disease-specific medications) or vaccine (including over the counter prescription medicines, recreational drugs, vitamins, and/or herbal supplements) that the participant had received within 2 months before triptorelin administration or receives during the study must be recorded on the eCRF along with:

- Generic or trade name
- Reason for use
- Dates of administration including start and end dates
- Dosage information including dose, frequency and route of administration

The medical monitor should be contacted if there are any questions regarding concomitant or prior therapy.

The following concomitant medications are not permitted during this study:

- Any treatment or procedure with a specific or potential effect on androgenic hormones be administered concomitantly to the study drug (will be considered as a protocol violation). Per investigator's clinical judgement, suggest offering short-term administration of an older generation androgen receptor antagonist to M1 participants starting study intervention to reduce the risk of the 'flare-up' phenomenon.
- Any medication which raises prolactin levels and those affecting pituitary secretion of gonadotropins
- All drugs mentioned as prohibited in the exclusion criteria:
  - o Finasteride or dutasteride.
  - o Medications which are known to affect the metabolism and/or secretion of androgenic hormones: ketoconazole, aminoglutethimide, oestrogens.
  - o Systemic or inhaled corticosteroids (topical application permitted).
  - o Cytotoxic chemotherapy, abiraterone.
  - o Any traditional Chinese medicine or herbal products previous used within 1 month prior to study start or plan to be used during the study, which are known to have cytotoxic effect or affect the metabolism and/or secretion of androgenic hormones.
  - o Concomitant use of medications known to prolong QT interval should not be given (class IA (e.g. quinidine, disopyramide) or class III (e.g. amiodarone, sotalol, dofetilide, ibutilide) antiarrhythmic medicinal products, methadone, moxifloxacin, antipsychotics).

The following concomitant medications are permitted during this study, but they must be monitored closely, and every effort should be made to keep their dose and dose regimen constant throughout the course of the study:

- Analgesics: are allowed when necessary for pain relief.
- Anticonvulsants (e.g phenobarbital): long-term therapy may have additional risk for osteoporosis.
- Other medications: any treatment which is considered necessary for the participant's welfare, may be given at the discretion of the investigator.

IPSEN GROUP D-CN-52014-237

CONFIDENTIAL PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024


Other procedures: any diagnostic, therapeutic or surgical procedure performed during the study period should be recorded, including the date, indication, description of the procedure(s), and any clinical findings.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 39/92

# 7 DISCONTINUATION OF STUDY INTERVENTION AND PARTICIPANT DISCONTINUATION/WITHDRAWAL

Discontinuation of specific sites or of the study as a whole are detailed in Section 10.1.8.

#### 7.1 Discontinuation of Study Intervention

In this study, there will only be one treatment cycle administered on Day 1 of the study, thus discontinuation of the study intervention is not applicable (i.e. no repeat cycles). In the event a participant is enrolled, but does not receive study intervention, the participant will not remain in the study and EoS/EW assessment will not be performed. Only the reason for discontinuation will be collected.

If participants are lost to follow-up, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.

#### 7.1.1 Temporary Discontinuation

In case of suspected or confirmed COVID-19 (SARS-CoV-2) infection, the intervention administration may be temporarily postponed depending on the participant clinical presentation. In some cases, the investigator may request a participant be retested before the intervention administration.

# 7.2 Participant Discontinuation/Withdrawal from the Study

- A participant may withdraw from the study at any time at his/her own request or may be withdrawn at any time at the discretion of the investigator for safety, behavioural or compliance reasons.
- At the time of discontinuing from the study, an early discontinuation visit should be conducted, as shown in the SoA. See SoA for data to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed.
- The reason for discontinuation will be recorded in the eCRF.
- If the participant withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such withdrawal of consent.
- If the participant withdraws consent for any further contact, the investigator will explain in the medical records that the participant was also withdrawn from study procedures. This information must be entered in the eCRF.
- If a participant withdraws from the study, he/she may request destruction of any samples taken and not tested, and the investigator must document this in the site study records.
- A participant will be withdrawn from the study if they have inadequate testosterone suppression (defined as >50 ng/dL detected at least 30 days after administration of study intervention and on two consecutive measurements at least 2 weeks apart, at either a scheduled or unscheduled study visit).

# 7.3 Lost to Follow-up

A participant will be considered lost to follow-up if they repeatedly fail to return for scheduled visits and is unable to be contacted by the study site.

The following actions must be taken if a participant fails to return to the clinic for a required study visit:

• The site must attempt to contact the participant and reschedule the missed visit as soon as possible. The site should counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether the participant wishes to and/or should continue in the study.

# IPSEN GROUP D-CN-52014-237


# CONFIDENTIAL PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024

• Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, three telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record.

- Should the participant continue to be unreachable, he/she will be considered to have withdrawn from the study.
- Site personnel will attempt to collect the vital status of the participant within legal and ethical boundaries for all participants enrolled, including those who did not receive study intervention. Public sources may be searched for vital status information. If vital status is determined as deceased, this will be documented, and the participant will not be considered lost to follow-up. Sponsor personnel will not be involved in any attempts to collect vital status information.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 41/92

#### 8 STUDY ASSESSMENTS AND PROCEDURES

- Study procedures and their timing are summarised in the SoA (Table 1 and Table 2). Protocol waivers and exemptions are not allowed.
- Immediate safety concerns should be discussed with the sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue study intervention.
- Adherence to the study design requirements, including those specified in the SoA (Table 1 and Table 2), is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.
- Procedures conducted as part of the participant's routine clinical management (e.g. blood count) and obtained before signing of the ICF may be utilised for screening or baseline purposes provided the procedures met the protocol-specified criteria and were performed within the timeframe defined in the SoA (Table 1 and Table 2)
- The maximum amount of blood collected from each participant over the duration of the study, including any extra assessments that may be required, will not exceed 95 mL for the PK/PD subset of participants and 60 mL for all other participants. Blood sampling should be taken at the same time of day during different visits.
- Repeat or unscheduled samples may be taken for safety reasons or in case of technical issues with the samples.

#### 8.1 Demography

Age, sex and, according to individual country regulations/requirements and if authorised in the country, race/ethnicity will be collected.

#### 8.2 Efficacy Assessments

Efficacy will be assessed in this study using the surrogate PD markers for testosterone and PSA concentrations.

Approximately 26 mL of blood will be collected from all participants, and approximately 38 mL of blood from the PK/PD subset participants, for measurement of testosterone and PSA. Serum samples used to evaluate testosterone and PSA will be divided into two aliquots (one primary and one back-up).

Further instructions for the collection, handling and shipment of biological samples will be provided by the sponsor and described in the study Laboratory Manual.

### 8.2.1 Testosterone

Testosterone will be assessed by a third-party vendor, as described in the Laboratory Manual. Serum will be analysed to determine concentrations of testosterone using a validated, specific and sensitive liquid chromatography tandem mass spectrometry (LC-MS/MS) methods.

Blood samples for the determination of testosterone serum concentrations will be collected at the timepoints indicated in the SoA (Table 1 (all participants) and Table 2 (for the subset of 12 participants)).

Residual serum samples remaining from the analysis may also be retained by the sponsor for up to 5 years after completion of the study. This could include using leftover serum for long-term stability or reproducibility assessments.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 42/92

Surplus serum samples can only be used in China. Surplus serum samples will be managed anonymously and will not be identifiable.

#### 8.2.2 Prostate-specific Antigen

PSA will be assessed centrally, as described in the study Laboratory Manual.

Blood samples for the determination of PSA plasma concentrations will be collected at the timepoints indicated in Table 1 (all participants) and Table 2 (for the subset of 12 participants).

### 8.3 Safety Assessments

Planned time points for all safety assessments are provided in the SoA. Evaluations obtained as part of routine medical care and performed during the screening period may be used in place of the study specific evaluations. Participants will acknowledge and agree to the possible use of this information for the study by giving informed consent.

#### 8.3.1 Physical Examinations

A complete physical examination will include, at a minimum, assessments of the skin, and cardiovascular, respiratory, gastrointestinal and neurological systems. Height and weight will also be measured and recorded. Body weight will be measured in underwear and without shoes.

A brief physical examination will include, at a minimum, assessments of the lungs, cardiovascular system, abdomen (liver and spleen).

Investigators should pay special attention to clinical signs related to previous serious illnesses. Any clinically significant physical examination findings (abnormalities) observed during the study will be reported as AEs. Any physical examination findings (abnormalities) persisting at the end of the study will be followed by the investigator until resolution or until clinically stable. In addition, participants, particularly those with M1b status, should be advised regarding clinical signs suggestive of spinal cord compression.

#### 8.3.2 Vital Signs

Blood pressure, temperature, respiratory rate and heart rate will be assessed as outlined in the SoA (Section 1.3) with an automated device (if possible) so that measurements are independent of the observer. Blood pressure and heart rate will be recorded after 5 minutes rest in supine or seated position. Absolute values and change from Baseline will be analysed. Any clinically significant vital signs will be recorded as AEs.

## 8.3.3 Electrocardiograms

A 12-lead ECG analysis will be included as a safety evaluation/endpoint in this study at timepoints described in Table 1 and Table 2.

A single 12-lead ECG will be recorded so that the different ECG intervals (RR, PR, QRS, QT, QTcF) can be measured automatically. The ECG will be recorded with the participant in supine position after five minutes of rest until four regular consecutive complexes are available.

Any clinically significant abnormalities will be recorded as AEs.

#### 8.3.4 Magnetic Resonance Imaging Scan

A magnetic resonance imaging (MRI) scan for prostate gland or the whole body, only if necessary (based on investigator's judgement), will be performed as described in the SoA (Table 1 and Table 2) to confirm disease stage prior to study entry. An MRI scan is not required, if performed within 1 month of study screening.

#### 8.3.5 Clinical Safety Laboratory Assessments

- All clinical laboratory safety tests (haematology and blood biochemistry) will be assessed locally.
- See Appendix 10.2 for the list of clinical laboratory tests to be performed and to the SoA (Section 1.3) for the timing and frequency.
- The investigator must review the laboratory report, document this review, and record any clinically significant changes occurring during the study as an AE. The laboratory reports must be filed with the source documents.
- Abnormal laboratory findings associated with the underlying disease, are not considered clinically significant unless judged by the investigator to be more severe than expected for the participant's condition.
- All laboratory tests with values considered clinically significantly abnormal during participation in the study or within 168 days after the last dose of study intervention should be repeated until the values return to normal or baseline or are no longer considered clinically significant by the investigator or medical monitor.
  - If clinically significant values do not return to normal/baseline within a period of time judged reasonable by the investigator, the aetiology should be identified, and the sponsor notified.
  - All protocol-required laboratory tests, as defined in Appendix 10.2, must be conducted in accordance with the laboratory manual and the SoA (Section 1.3).
  - If laboratory values from non-protocol specified laboratory tests performed at the study site laboratory require a change in participant management or are considered clinically significant by the investigator (e.g. SAE or AE or dose modification), then the results must be recorded in the eCRF.

Haematology blood samples (2 mL) will be collected in a potassium ethylenediaminetetraacetic acid tube. Blood biochemistry samples (3 mL) will be collected in an activator gel tube.

#### 8.3.6 Local Tolerance

Local tolerance will be assessed 2 hours ( $\pm 15$  minutes) after injection. After the single injection of 6-month formulation triptorelin, the injection site will be examined by a physician or Medical Research Associate and assessed for characteristics such as but not limited to tenderness, redness, bruising, erythema, swelling, rash, pain, itching, induration, haematoma, ulceration or necrosis. If present, the extent of erythema, haematoma, rash, ulceration or necrosis will be described and assessed quantitatively; this will at least include measurement of maximum length and maximum width. If any reactions meet the definition of a treatment-emergent adverse event (TEAE), they are to be reported in the eCRF as such (see Section 9.4.5).

# 8.4 Adverse Events (AEs) and Serious Adverse Events (SAEs), and Other Safety Reporting

The definitions of AEs and serious adverse events (SAEs) can be found in Appendix 10.3. Adverse events will be reported by the participant (or, when appropriate, by a caregiver, surrogate).

The investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible for following up all AEs or SAEs, considered related to the study intervention or study procedures (see Section 7).

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 44/92

The method of recording, evaluating, and assessing causality of AEs and SAEs and the procedures for completing and transmitting SAE reports are provided in Appendix 10.3.

# 8.4.1 Time Period and Frequency for Collecting AE and SAE Information

All AEs and SAEs will be collected from the signing of the ICF until the EoS at the time points specified in the SoA (Section 1.3).

Medical occurrences that begin before the start of study intervention but after obtaining informed consent will be recorded on the AE section of the case report form.

All SAEs will be recorded and reported to the sponsor or designee immediately and under no circumstance should this exceed 24 hours of awareness of the event, as indicated in Appendix 10.3. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.

Investigators are not obligated to actively seek information on AEs or SAEs after conclusion of the study participation. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event to be reasonably related to the study intervention or study participation, the investigator must promptly notify the sponsor.

#### 8.4.2 Method of Detecting AEs and SAEs

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the participant is the preferred method to inquire about AE occurrences.

## 8.4.3 Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All AEs/SAEs will be followed until resolution or stabilisation or the participant is lost to follow-up (as defined in Section 7.3). Further information on follow-up procedures is provided in Appendix 10.3.

#### 8.4.4 Regulatory Reporting Requirements for SAEs

- Prompt notification by the investigator to the sponsor of an SAE is essential so that legal obligations and ethical responsibilities towards the safety of participants and the safety of a study intervention under clinical investigation are met.
- The sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a study intervention under clinical investigation. The sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, Institutional Review Boards (IRB)/Independent Ethics Committees (IEC), and investigators.
- An investigator who receives an investigator safety report describing an SAE or other specific safety information (e.g. summary or listing of SAEs) from the sponsor will review and then file it along with the Investigator's Brochure and will notify the IRB/IEC, if appropriate according to local requirements.
- Investigator safety reports must be prepared for suspected unexpected serious adverse reactions (SUSAR) according to local regulatory requirements and sponsor's policy and forwarded to investigators as necessary.

#### 8.4.5 Pregnancy

All participants in this study are male. The investigator must instruct all male participants to inform the investigator immediately should their partner become pregnant.

- Details of all pregnancies in female partners of male participants will be collected from the signing of the ICF and until up to 9 months after the participants last dose of study intervention.
- If a pregnancy is reported, the investigator will record pregnancy information on the appropriate forms (Pregnancy Notification Form- paper form) and submit it to the sponsor within 24 hours of learning of the female partner of male participant becoming pregnant (after obtaining the necessary signed informed consent from the female partner).
- Any pregnancy complication or elective termination of a pregnancy for medical reasons will be reported as an AE or SAE.
- Abnormal pregnancy outcomes (e.g. spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs and will be reported as such.
- The participant's pregnant female partner will be followed to determine the outcome of the pregnancy unless consent is not given/withdrawn. The investigator will collect follow-up information on the participant's pregnant female partner and the neonate and the information will be forwarded to the sponsor.
- Any post-study pregnancy-related SAE considered reasonably related to the study intervention by the investigator will be reported to the sponsor as described in Section 8.4.4. While the investigator is not obligated to actively seek this information in a former study participant's pregnant female partner, he or she may learn of an SAE through spontaneous reporting.

#### 8.4.6 Disease-Related Events and/or Disease-Related Outcomes Not Qualifying as AEs or SAEs

Not applicable.

#### **8.4.**7 Adverse Events of Special Interest

Not applicable.

#### 8.4.8 Reporting of Study Intervention Errors Including Misuse/Abuse

- Medication errors are unintentional errors in the prescribing, storing, dispensing, preparing or administration of a study intervention (medicinal product) while under the control of a healthcare professional, participant or consumer.
- Misuse refers to situations where the study intervention is intentionally and inappropriately used not in accordance with the protocol.
- Abuse corresponds to the persistent or sporadic, intentional excessive use of a medicinal product, which is accompanied by harmful physical or psychological effects.
- Study intervention errors and uses outside of what is foreseen in the protocol will be recorded in the eCRF irrespective of whether associated with an AE/SAE or not. It will also be documented in the AE section of the eCRF if associated with an AE. It will be reported in the safety database only if associated with an SAE.

#### **Pharmacokinetics** 8.5

Approximately 14 mL of blood will be collected from all participants, and approximately 40 mL of blood from the PK/PD subset participants, for measurement of plasma concentrations of triptorelin 6-month formulation as specified in the SoA (Section 1.3)


# CONFIDENTIAL PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024

• Instructions for the collection, handling and shipment of biological samples will be provided by the sponsor and described in the study laboratory manual. The accurate date and time (24-hour clock time) of each sample collection must be recorded.

- Plasma samples will be used to evaluate the PK of triptorelin 6-month formulation. Each plasma sample will be divided into two aliquots (one primary and one backup). Samples collected for analyses of triptorelin concentration may also be used to evaluate safety or efficacy aspects related to concerns arising during or after the study.
- During the study, the nominal sample collection times may be changed, but the total number of samples will not increase. The exact dates and times of blood sample collection and study drug administration must be recorded in the eCRF.
- On predetermined dates, plasma samples will be shipped to the bioanalytical service provider under frozen conditions. For security reasons, the back-up aliquots will not be shipped until the primary aliquots have arrived. Upon receipt at the bioanalytical service provider, samples will be checked and stored until analysis.
- Plasma will be analysed to determine concentrations of triptorelin using a validated, specific and sensitive LC-MS/MS methods.
- Surplus plasma samples will be used in China and will not be shipped outside China. Surplus plasma samples will be managed anonymously and will not be identifiable.
- Residual plasma samples remaining from the analyses may also be retained by the sponsor for up to 5 years after completion of the study. This could include using leftover plasma for long-term stability or reproducibility assessments.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 47/92

#### 9 STATISTICAL CONSIDERATIONS

#### 9.1 Statistical Hypotheses

No statistical hypotheses are planned for this study.

# 9.2 Sample Size Determination

The sample size was estimated based on data from the previous Study DEB-TRI6M-301, 97.5% of participants achieving castration and 93% of participants maintaining castration from Week 8 to Week 24.

Sample size is calculated to fulfil the co-primary efficacy criteria of this study, which is to assess the proportion of participants achieving castrate levels of testosterone on Day 29 and the proportion of participants maintaining the castrate levels of serum testosterone from Week 8 to end of Week 24. A total of 195 participants with advanced prostate cancer will be enrolled to receive the triptorelin pamoate 22.5 mg 6-month formulation.

For an exact binomial test of a proportion with a two-sided nominal significance level of 0.05 and null proportion of 85%, a sample size of 165 participants has an exact power of 88.3% when the true proportion is 93% (of participants maintaining castration from Week 8 to Week 24). This sample size of 165 participants has a power >99.9% when the true proportion is 97.5% (of participants achieving castrate testosterone levels). Exact two-sided 95% confidence interval (CI) for a binomial proportion was computed by SAS using the exact binomial distributions.

Assuming the dropout rate will be around 15%, a sample size of 195 participants in total is planned for this study.

## 9.3 Analysis Sets

For the purposes of analysis, the following analysis sets are defined:

| Participant Analysis Set | Description |
|---|---|
| Screened | All participants screened (i.e. who signed the informed consent). |
| Safety Set | The safety set will contain all participants who receive the single dose of study intervention. |
| Full Analysis Set | The FAS will contain all treated participants who complete the study or is a treatment failure. |
| | Completing the study is defined as having serum testosterone measurement at baseline, Day 29 and Day 169. Treatment failure is defined as escaping castration (testosterone level ≥50 ng/dL) at any assessments on and after Day 29 during the study, or premature discontinuation from the intervention period due to drug-related reasons (adverse event or death). |
| Per Protocol Set | All participants in the FAS who have no impacting major protocol deviations (i.e. that could potentially affect the primary efficacy endpoint outcome for the participant) as described in the protocol deviations document. |
| Rich PK Analysis set (for non-compartmental analysis) | Participants in the PK/PD subset who receive one dose of study intervention, have no major protocol deviations affecting the PK variables, and who have a sufficient number of plasma concentrations to estimate the main PK parameters (maximum observed plasma drug concentration ( $C_{max}$ ), time to maximum observed drug concentration ( $t_{max}$ ) and area under the plasma concentration time curve (AUC)) |
| Population PK Analysis Set | All participants who received one dose of triptorelin and who have at least one triptorelin plasma concentration and no major protocol deviations affecting PK variables. |

# CONFIDENTIAL

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 48/92

| Participant Analysis Set | Description |
|---|---|
| Rich PD Analysis Set | all participants in the PK/PD subset who have a sufficient number of PD (testosterone) measurements to estimate the main PD parameters (maximum observed concentration ( $C_{max}$ ), time to maximum observed concentration ( $t_{max}$ ) and time to castration ( $t_{cast}$ )) |

FAS=full analysis set; PD=pharmacodynamic PK=pharmacokinetic

The efficacy analysis for the primary and secondary efficacy endpoints will be presented for the full analysis set (FAS) and per protocol (PP) population. The analysis of the safety data will be performed based on the safety set and analysis of PK and PD in the relevant PK analysis set

#### 9.4 Statistical Analyses

The statistical analysis plan (SAP) will be finalised before the first participant enters the study and it will include a more technical and detailed description of the statistical analyses described in this section. This section is a summary of the planned statistical analyses of the most important endpoints including primary and key secondary endpoints.

Other endpoints as well as demographic, baseline characteristics and disposition will be detailed in the SAP.

Statistical evaluation will be performed using Statistical Analysis System (SAS®) Version 9.4 (or higher if available).

#### 9.4.1 General Considerations

#### 9.4.1.1 Reasons for Exclusion from the Analyses

Any major protocol deviation will be described and listed and its impact on inclusion of any participant in each analysis population will be specified. The final list of protocol deviations impacting each analysis population will be reviewed prior to database lock. The list may be updated, up to the point of database lock, to include any additional major protocol deviations impacting inclusion in the PP set.

#### 9.4.1.2 Significance Testing and Estimations

As this is a descriptive safety and efficacy study, no formal statistical testing will be carried out.

#### 9.4.1.3 Statistical/Analytical Methods

Statistical analyses will be performed by an external CRO, managed by the sponsor's Biometry department.

# Demographic and Other Baseline Characteristics

Descriptive summary statistics (n, mean, standard deviation (SD), median, minimum, maximum) or frequency counts of demographic and baseline data (medical history, concomitant disease (predosing AEs and ongoing medical history, prior medications and therapies, etc.) will be presented for the FAS, PP and safety sets.

#### Participant Disposition and Withdrawals

The numbers and percentages of participants screened and included in each of the populations will be tabulated overall and by centre. The reasons for participant exclusions from each of the populations will also be tabulated. Primary reasons for discontinuation of study will be tabulated.

### Adjustment for Country/Centre Effects

Descriptive analysis will be carried out to evaluate any possible centre effect.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 49/92

### 9.4.2 Analysis of Primary Endpoints

The co-primary efficacy variables are

- percentage of participants achieving castrate levels of serum testosterone (<50 ng/dL or 1.735 nmol/L) and
- percentage of participants maintaining the castrate levels from Week 8 to Week 24.

The percentage of participants achieving castrate levels of serum testosterone (<50 ng/dL or 1.735 nmol/L) on Day 29 will be obtained as the number of participants with castrate levels at the visit, divided by the total number of participants on Day 29 in the considered population.

Percentage of participants maintaining the castrate levels of serum testosterone (<50 ng/dL or 1.735 nmol/L) from Week 8 to Week 24 will be calculated as the number of participants with castrate levels at all visits from Week 8 to Week 24, divided by the total number of assessable participants.

To derive the percentage of participants maintaining castration levels of testosterone, missing data will be handled as follows:

- (a) In participants escaping castration at a certain visit, subsequent missing data is irrelevant.
- (b) Participants maintaining castration up to a certain visit with missing data afterwards (drop-out due to non-drug-related reasons) will be excluded from the analysis.
- (c) Participants maintaining castration up to a certain visit with missing data afterwards (drop-out due to drug-related reasons) will be treated as having escaped castration (failure).
- (d) Missing data between two visits where castration levels are maintained will be handled as missing for that particular visit, and the participant will be considered to have maintained castration.

To derive the percentage of participants maintaining castrate levels of testosterone, assessable participants are defined as the total number of all participants having values at all visits and all participants having missing data according to the criteria a), c) and d) mentioned previously. Participants having missing data according to the criteria b) will be excluded from this calculation.

Co-primary endpoints will be tabulated with two-sided 95% (95% CI) using the Clopper-Pearson exact method.

### 9.4.3 Analysis of Secondary Endpoints

#### 9.4.3.1 Prostate-Specific Antigen

The secondary efficacy variable is the percent change in PSA from baseline (prior to injection) measured at Week 12 and Week 24. Percent change in PSA is defined as the absolute value of difference between the PSA values at Week 12 and Week 24 and the baseline value divided by the baseline value.

PSA percent change from pre-treatment Day 1 will be reported at each subsequent visit, using descriptive statistics.

### 9.4.3.2 Pharmacokinetic and Pharmacodynamic Data Analysis

#### Description of Triptorelin and Testosterone Concentrations

Individual plasma or serum concentrations of triptorelin and testosterone will be listed and summarised by visit and time points using descriptive statistics for continuous variables (number of available observations, mean, median, SD, minimum, maximum, geometric mean, and geometric coefficient of variation (assuming log normally distributed data). Data will be

summarised for the PK/PD subset and overall. Individual and mean triptorelin and testosterone concentration time profiles, as well as spaghetti plots, will be generated.

#### Non-compartmental Analysis

The PK analysis of triptorelin plasma concentrations and testosterone serum concentrations of the rich sampling PK/PD subset will be performed by the non-compartmental analysis (NCA) approach using Phoenix WinNonlin PK program version 8.3 or higher. The following PK parameters will be calculated if warranted by the data:

- maximum observed concentration (C<sub>max</sub>)
- time to maximum observed blood concentration  $(t_{max})$
- (for triptorelin only) area under the plasma concentration time curve from time 0 to the time of the last quantifiable concentration (AUC<sub>last</sub>)
- (for triptorelin only) area under the plasma concentration time curve from time 0 to the visit on day  $169 \text{ (AUC}_{0-169})$
- (For testosterone only): time to castration t<sub>cast</sub>

Additional PK parameters may be calculated if appropriate.

Descriptive statistics of PK and PD parameters will be presented for the rich PK analysis set for triptorelin and the rich PD analysis set for testosterone. PK and PD parameters will be summarised by, but not limited to, n, mean, SD, median, minimum, maximum, geometric SD, geometric mean, and geometric coefficient of variation except for  $t_{max}$  where only n, median, minimum and maximum values will be reported.

The NCA analysis will be described in a separate data analysis plan and reported in a standalone report.

#### Population Pharmacokinetic Analysis

Population pharmacokinetics (PopPK) modelling will be performed using concentrations obtained from all participants in order to describe the pharmacokinetics of triptorelin 6-month formulation in the prostate cancer population (if warranted by the data). In addition, quantification of the inter-participant variability on PK will be performed and an attempt to identify participant characteristics explaining the variability on PK will be made. Historical PK data from other studies may also be used to compare the PK profiles from this study against other populations. The PK model developed will be used to derive exposure metrics to perform an exploratory analysis with efficacy and safety endpoints (should any safety signal emerge). Should a trend be observed, PK/PD modelling will be performed to describe the relationship between exposure and efficacy and/or safety endpoints.

Population PK/PD analysis will be described in a separate data analysis plan and presented in a stand-alone report.

#### 9.4.4 Analysis of Exploratory Endpoint

#### 9.4.4.1 Pharmacokinetic/Pharmacodynamic Relationship

An exploratory analysis will be performed to assess the relationship between PK and PD endpoints. If a trend is shown, an attempt to build a PK/PD model using a population approach will be performed. The PopPK and PK/PD analyses will be described in a separate data analysis plan and reported in a standalone report.

#### 9.4.5 Safety Analyses

Safety endpoints are indicated in Section 3.

All safety data will be included in the participant data listings. Analyses and summary tables will be based upon the safety set.

All AEs will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) version 24.1 (or higher if available) and will be classified by MedDRA preferred term and system organ class. Adverse event listings will be presented by participant, system organ class and PT.

The incidence of all TEAEs and SAEs will be tabulated overall. In addition, summary tables will be presented by maximum intensity and drug relationship.

A TEAE is defined as any AE that occurs during the active phase of the study (from study intervention injection to 24 weeks after injection) if it was not present prior to receiving study intervention, or:

- it was present prior to receiving IMP but the intensity increased during the active phase of the study.
- It became serious during the active phase of the study
- It was present prior to receiving the study intervention and the intensity was the same, but the causality changed to 'related to treatment' during the active phase of the study.

All TEAEs will be flagged in the AEs listings.

Haematological and biochemical toxicities will be recorded and graded according to the NCI CTCAE criteria, where available. The National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Grade 3 and 4 haematology and biochemistry variables by participant and by cycle will be listed.

Actual values and changes from baseline in clinical laboratory tests, physical examinations, vital signs and 12-lead ECG will be summarized using descriptive statistics at each visit. For laboratory data, abnormal values will be flagged in the data listings and a list of clinically significant abnormal values will be presented. Shift tables using the worst on-treatment grade will be presented for the number and percentage of participants with NCI-CTCAE grades.

AEs reported by investigators using the NCI-CTCAE classification (Version 5.0 or higher) will be coded using MedDRA Version 24.1 (or higher if available).

Summary incidence tables will be provided, classified by SOC, PT and associated NCI/CTC worst grade. In the event of multiple occurrences of the same AEs being reported by the same participant, the maximum intensity (Grade 5 > Grade 4 > Grade 3 > Grade 2 > Grade 1 > missing > not applicable) will be chosen.

#### 9.4.6 Subgroups Analyses

No subgroups analysis will be performed.

#### 9.4.7 Other Analyses

Not applicable.

# 9.5 Interim Analyses

No interim analysis will be performed.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 52/92

# 10 SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

#### 10.1 Appendix: Regulatory, Ethical, and Study Oversight Considerations

## 10.1.1 Regulatory and Ethical Considerations

- This study will be conducted in accordance with the protocol and with the following:
  - Consensus ethical principles derived from international guidelines including the Declaration of Helsinki and Council for International Organisations of Medical Sciences International Ethical Guidelines
  - International Council for Harmonisation (ICH) Good Clinical Practice (GCP) Guidelines
  - Applicable laws and regulations such as Regulation EU 536/2014
- The protocol, protocol amendments, ICF, Investigator Brochure, and other relevant documents (e.g. any participant recruitment materials) must be approved by the IRB/IEC before the study is initiated.
- Any amendments to the protocol will require IRB/IEC approval before implementation of changes made to the study design, except for changes necessary to eliminate an immediate hazard to study participants.
- The protocol and any substantial amendments to the protocol will require health authority approval prior to initiation except for changes necessary to eliminate an immediate hazard to study participants.
- The investigator will be responsible for the following:
  - Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies, and procedures established by the IRB/IEC
  - Notifying the IRB/IEC of SAEs or other significant safety findings as required by IRB/IEC procedures
  - Providing oversight of the conduct of the study at the site and adherence to applicable local regulations, ICH guidelines and the IRB/IEC requirements/procedures.

#### 10.1.2 Financial Disclosure

Investigators and sub-investigators will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for one year after completion of the study.

## 10.1.3 Informed Consent Process

- The ICF and any participant recruitment materials must be in compliance with ICH GCP, local regulatory requirements, and legal requirements, including applicable privacy laws. They must be approved prior to use as described in Section 10.1.1.
- The investigator or his/her authorised representative will explain to the participant or their legally authorised representative the nature and objectives of the study and possible risks and benefits associated with the participation. They will answer all questions regarding the study.

- Participants or their legally authorised representative, when applicable must be informed that their participation is voluntary.
- The investigator or his/her authorised representative will obtain written informed consent from each participant or the legally authorised representative, when applicable, before any study-specific procedure is performed. The investigator will retain the original of each participant's signed ICF.
- A copy of the signed ICF(s) must be provided to the participant or their legally authorised representative.
- The medical record must include a statement that written informed consent was obtained before the participant was enrolled in the study and the date the written consent was obtained. The authorised person obtaining the informed consent must also sign the ICF.
- Participants must be re-consented to the most current version of the ICF(s) during their participation in the study. If changes to the ICF do not apply to all participants, this will be communicated to the IRB/IEC with a rationale. IRB/IEC approval must be received before implementation as required by local regulations.
- The ICF will contain a separate section that addresses the use of all data combined with data from prostate cancer patients from other parts of the world. These data may only be used for analysis to advance science and public health, including in order to:
  - understand and evaluate the study drug and/or other drugs,
  - better understand the studied disease and associated health problems,
  - develop new drugs and find new ways to detect, treat, prevent or cure health problems,
  - plan new studies or improve scientific analysis methods,
  - publish research results in scientific journals or use them for educational purposes,
  - conduct additional statistical analysis.
- Participants will be told that they are free to refuse to participate and may withdraw their consent at any time and for any reason during the study.
- If a pregnancy is reported for a female partner of a male participant during the study, the partner will be asked to sign appropriate consent for the sponsor to follow the outcome of the pregnancy.

#### 10.1.4 Data Protection

- Participants will be assigned a unique identifier by the sponsor. Any participant records or datasets that are transferred to the sponsor will contain the identifier only; participant names or any information which would make the participant identifiable will not be transferred.
- The participant must be informed that his/her personal study-related data will be used by the sponsor in accordance with local data protection law. The level of disclosure must also be explained to the participant who will be required to give consent for their data to be used as described in the informed consent.
- The participant must be informed that his/her medical records may be examined by the sponsor's auditors or other authorised personnel appointed by the sponsor, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.
- The sponsor will ensure that appropriate organisational and technical arrangements are implemented to comply with the applicable rules on the protection of personal data. In the event of a potential data security breach concerning personal data processed on behalf

of the sponsor, the data protection officer must be informed without undue delay and no later than 24 hours from the discovery of the event. The data protection officer will evaluate the event and notify the Data Protection Authorities within 72 hours, if required. Corrective actions and preventive actions will be implemented to mitigate the possible adverse effects. Affected study participants will be informed accordingly. Ipsen Data Protection Officer can be contacted by email: dataprivacy@ipsen.com.

• When permitted by local regulation, the ICF will contain a separate section that addresses the remote access by the study monitors to source documents/data for the purpose of source data verification. A specific consent will be required to document a participant's agreement.

# 10.1.5 Dissemination of Clinical Study Data

- The sponsor seeks to publish the results of its clinical trials in biomedical journals, whatever the outcome. Clinical trial results may also be presented at international congresses as posters or oral presentations.
- Protocol and result summary will be made publicly available on the US Clinical Trials Registry (ClinicalTrials.gov). The sponsor also provides clinical trial information to other national clinical trial registries or databases according to local requirements/legislation.
- A clinical study report will be prepared if at least one participant has signed informed consent and received intervention, regardless of whether the study is completed or prematurely terminated. The clinical study report may be disclosed according to regulatory requirements.

#### 10.1.6 Data Quality Assurance

- All participant data relating to the study will be recorded in the CRF unless transmitted to the sponsor or designee electronically (e.g. laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by signing the CRF.
- All entries in the CRF will be made under the e-signature of the person performing the action. This electronic signature consists of an individual and confidential username and password combination. It is declared to be the legally binding equivalent of the handwritten signature. Only sponsor authorised users will have access to the CRF as appropriate to their study responsibilities. Users must have successfully undergone software application training prior to entering data into the CRF.
- Guidance on completion of CRFs will be provided in CRF completion guidelines.
- The investigator must permit study-related monitoring, audits, IRB/IEC review, and regulatory authority inspections, and provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing, and inspection by domestic and foreign regulatory authorities.
- Monitoring details describing strategy, including definition of study critical data items and processes (e.g. risk-based initiatives in operations and quality such as Risk Management and Mitigation Strategies and Analytical Risk-Based Monitoring), methods, responsibilities and requirements, including handling of noncompliance issues and monitoring techniques (central, remote, or on-site monitoring) are provided in the Monitoring Plan.
- The sponsor or designee is responsible for the data management of this study including quality checking of the data.

- The sponsor assumes accountability for actions delegated to other individuals (e.g. Contract Research Organisations).
- Records and documents, including signed ICFs, pertaining to the conduct of this study should be retained by the investigator according to the ICH-GCP guidelines, to local regulations, or as specified in the study agreement, whichever is longer. No records may be destroyed during the retention period without the written approval of the sponsor. No records may be transferred to another location or party without written notification to the sponsor.

#### 10.1.7 Source Documents

- Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.
- Data reported in the CRF that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.
- Definition of what constitutes source documents/data and their location will be documented in a specific form.
- The investigator must maintain accurate documentation that supports the information entered in the CRF. Source data must be attributable, legible, contemporaneous, original, accurate and complete.
- Study monitors will perform ongoing source data verification to confirm that data entered into the CRF by authorised site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements. When permitted by local regulation and guidance, study monitors will access remotely to source documents/data to conduct source data verification, while maintaining appropriate security measures and ensuring the protection of the data. This will be described in the monitoring plan or equivalent.

#### 10.1.8 Study and Site Start and Closure

#### First Act of Recruitment

The study start date is the date on which the clinical study will be open for recruitment of participants or the actual date on which the first participant is enrolled.

# **Study/Site Termination**

There are no formal rules for early termination of this study.

The sponsor or designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of the sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

For study termination:

• Discontinuation of further study intervention development


For site termination:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate or no recruitment (evaluated after a reasonable amount of time) of participants by the investigator
- Total number of participants included earlier than expected

If the study is prematurely terminated or suspended, the sponsor shall promptly inform the investigators, the IECs/IRBs, the regulatory authorities, and any contract research organization(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements. The investigator shall promptly inform the participant and should assure appropriate participant therapy and/or follow-up.

# 10.1.9 Publication Policy

- The results of this study may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.
- The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multicentre studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement.
- Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.


PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 57/92

### **10.2** Appendix: Clinical Laboratory Tests

- The tests detailed in Table 6 will be performed locally.
- Protocol-specific requirements for inclusion or exclusion of participants are detailed in Section 5 of the protocol.
- Additional tests may be performed at any time during the study as determined necessary by the investigator or required by local regulations.
- Refer to SoA Section 1.3 for details of visits.

Table 6 Protocol-Required Safety Laboratory Tests

| Parameters | Screening | Intervention Period | EoS/EW |
|---|---|---|---|
| Haematology | X | X | X |
| Platelet Count | X | X | X |
| Haemoglobin | X | X | X |
| White blood cell count with differential:<br>Neutrophils | X | X | X |
| Lymphocytes | | | |
| Monocytes | | | |
| Eosinophils | | | |
| Basophils | | | |
| Clinical Chemistry | | | |
| Creatinine | X | X | X |
| Glucose (fasted at screening and fasted on Day 1 and Day 169) [a] | X | X | X |
| Aspartate aminotransferase | X | X | X |
| Alanine aminotransferase | X | X | X |
| Alkaline phosphatase | X | X | X |
| Bilirubin (total and conjugated) | X | X | X |

EoS=end of study; EW=early withdrawal

Note: All parameters will be analysed locally. The preparation and storage of samples will be performed per each local laboratory practice.

Investigators must document their review of each laboratory safety report.

a Fasting not necessary for diabetic participants.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 58/92

# 10.3 Appendix: AEs and SAEs: Definitions and Procedures for Recording, Evaluating, Follow-up, and Reporting

#### 10.3.1 Definition of AE

#### **AE Definition**

- An AE is any untoward medical occurrence in a clinical study participant, temporally
  associated with the use of study intervention, whether or not considered related to the
  study intervention.
- NOTE: An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.

# Events Meeting the AE Definition

- Any abnormal laboratory test results (haematology, clinical chemistry, or urinalysis)
  or other safety assessments (e.g. ECG, radiological scans, vital signs measurements),
  including those that worsen from baseline, considered clinically significant in the
  medical and scientific judgment of the investigator (i.e. not related to progression of
  underlying disease).
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New condition detected or diagnosed after study intervention administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected intervention-intervention interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.
- "Lack of efficacy" or "failure of expected pharmacological action" per se will not be reported as an AE or SAE. Such instances will be captured in the efficacy assessments. However, the signs, symptoms, and/or clinical sequelae resulting from lack of efficacy will be reported as AE or SAE if they fulfil the definition of an AE or SAE.

#### Events NOT Meeting the AE Definition

- Any clinically significant abnormal laboratory findings or other abnormal safety
  assessments that are associated with the underlying disease, unless judged by the
  investigator to be more severe than expected for the participant's condition.
- The disease/disorder being studied or expected progression, signs or symptoms of the disease/disorder being studied, unless more severe than expected for the participant's condition.
- Medical or surgical procedure (e.g. endoscopy, appendectomy): the condition that leads to the procedure is the AE.

Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).


 Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

#### 10.3.2 Definition of SAE

An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed:

#### a. Results in death

#### b. Is life-threatening

The term 'life-threatening' in the definition of 'serious' refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

# c. Requires inpatient hospitalisation or prolongation of existing hospitalisation

In general, hospitalisation signifies that the participant has been admitted (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalisation are AEs. If a complication prolongs hospitalization or fulfils any other serious criteria, the event is serious. When in doubt as to whether "hospitalisation" occurred or was necessary, the AE should be considered serious.

Hospitalisation for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

#### d. Results in persistent or significant disability/incapacity

The term disability means a substantial disruption of a person's ability to conduct normal life functions.

This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhoea, influenza and accidental trauma (e.g. sprained ankle) that may interfere with or prevent everyday life functions but do not constitute a substantial disruption.

#### e. Is a congenital anomaly/birth defect

#### f. Other situations:

Medical or scientific judgment should be exercised by the investigator in deciding whether SAE reporting is appropriate in other situations such as significant medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These events should usually be considered serious.

Examples of such events include invasive or malignant cancers, intensive treatment for allergic bronchospasm, blood dyscrasias, convulsions or development of intervention dependency or intervention abuse.

A suspected or confirmed coronavirus COVID-19 (SARS-CoV-2) infection should be reported as serious if the event meets the defined seriousness criteria. If no seriousness criteria are reported by the investigator, the COVID-19 event will be collected and recorded as nonserious.

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 60/92

### 10.3.3 Recording and Follow-Up of AE and/or SAE

#### AE and SAE Recording

- When an AE/SAE occurs, it is the responsibility of the investigator to review all documentation (e.g. hospital progress notes, laboratory reports, and diagnostics reports) related to the event.
- The investigator will then record all relevant AE/SAE information.
- It is **not** acceptable for the investigator to send photocopies of the participant's medical records to the sponsor in lieu of completion of the required forms.
- There may be instances when copies of medical records for certain cases are requested
  by the sponsor. In this case, all participant identifiers, with the exception of the
  participant number, will be redacted on the copies of the medical records before
  submission to the sponsor.
- The investigator will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. Whenever possible, the diagnosis (not the individual signs/symptoms) will be documented as the AE/SAE.

#### Assessment of Intensity

The investigator will make an assessment of intensity for each AE and SAE reported during the study using the National Cancer Institute - Common Toxicity Criteria for AEs (NCI-CTCAE) Version 5.0 grading system.

#### Where:

- Grade 1: Mild; symptoms do not alter the participant's normal functioning.
- **Grade 2**: Moderate; symptoms produce some degree of impairment to function, but are not hazardous, uncomfortable or embarrassing to the participant.
- **Grade 3**: Severe; symptoms definitely hazardous to wellbeing or causing significant impairment of function or incapacitation.
- **Grade 4**: Life-threatening; any event that places the participant at immediate risk of death from the event as it occurred, i.e. it does not include a reaction that, had it occurred in a more severe form, might have caused death.
- Grade 5: Death related to AE

An event is defined as "serious" when it meets at least one of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

#### Assessment of Causality

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE/SAE. The investigator will use clinical judgment to determine the relationship.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration will be considered and investigated.

- The investigator will also consult the Investigator's Brochure (IB) and/or Product Information, for marketed products, in his/her assessment.
- For each AE/SAE, the investigator **must** document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred, and the investigator has
  minimal information to include in the initial report to the sponsor. However, it is very
  important that the investigator always make an assessment of causality for every event
  before the initial transmission of the SAE data to the sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

### Follow-up of AEs and SAEs

- The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by the sponsor to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.
- New or updated information will be recorded in the CRF.
- The investigator or qualified designee will submit any updated SAE data to the sponsor within 24 hours of receipt of the information.

#### 10.3.4 Reporting of SAEs

#### SAE Reporting to the sponsor via an Electronic Data Collection Tool

- The primary mechanism for reporting an SAE to the sponsor will be the electronic data collection tool.
- If the electronic system is unavailable, then the site will use the paper SAE data collection tool (see next section) to report the event within 24 hours of awareness of the event. The site will enter the SAE data into the electronic system as soon as it becomes available.
- After the study is completed at a given site, the electronic data collection tool will be taken off-line to prevent the entry of new data or changes to existing data.
- If a site receives a report of a new SAE from a study participant or receives updated data on a previously reported SAE after the electronic data collection tool has been taken off-line, then the site can report this information on a paper SAE form (see next section).
- Contacts for SAE reporting can be found on the SAE form and the cover sheet.

#### SAE Reporting to sponsor via paper

The site will email the SAE form or fax the cover sheet and SAE form to the sponsor
if the electronic data collection tool is unavailable. It must be retrospectively recorded
as soon as the electronic data collection tool becomes available.

# IPSEN GROUP D-CN-52014-237

CONFIDENTIAL PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024


• Contacts for SAE reporting can be found on the SAE form and the cover sheet.

# 10.4 Appendix: American Joint Committee on Cancer (AJCC) TNM Staging System for Prostate Cancer

The treatment of prostatic carcinoma is predicated largely on the stage of the disease; accurate staging is therefore essential.

The TNM staging system classifies the disease according to the progression of the primary tumour, the spread to the regional lymph nodes, and the development of distant metastases (hence TNM). Each stage is further subdivided (e.g. T1-T4 and Tla-T4) to give more detailed information about progression within each category.

| Primary Tumour (T) | T |
|---|---|
| Clinically inapparent tumour neither palpable nor visible by imaging: | T1 |
| Tumour incidental histologic finding in 5% or less of tissue resected | Tla |
| Tumour incidental histologic finding in more than 5% of tissue resected | Tl b |
| Tumour identified by needle biopsy (e.g. because of elevated PSA) | Tl c |
| Tumour confined within prostate | <b>T2</b> |
| Tumour found in one or both lobes by needle biopsy, but not palpable, or reliably visible | |
| by imaging is classified as TIc | |
| Tumour involves one half on one lobe or less | T2a |
| Tumour involves more than one half of one lobe but not both lobes | T2 b |
| Tumour involves both lobes | Т2 с |
| Tumour extends through the prostate capsule | Т3 |
| Invasion into the prostatic apex or into (but not beyond) the prostatic capsule is classified not as T3 but T2. | |
| Extracapsular extension (unilateral or bilateral) | T3a |
| Tumour invades seminal vesicles | T3b |
| Tumour is fixed or invades adjacent structures other than seminal | T4 |
| vesicles: bladder neck, external sphincter, rectum, levator muscles | 14 |
| and/or pelvic wall | |
| Regional Lymph Nodes (N) | N |
| No regional lymph node metastasis | NO |
| Metastasis in regional lymph node(s) | N1 |
| Distant metastasis (M) | M |
| No distant metastasis | MO |
| Distant metastasis | M1 |
| Non-regional lymph node(s) | Mla |
| Bone(s) | Mlh |
| Other site(s) with or without bone disease | Mlc |

# 10.5 Appendix: ECOG Performance Scale

These scales and criteria are used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis. They are included here for health care professionals to access.

| ECOG PERFORMANCE STATUS* | |
|---|---|
| Grade | ECOG |
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair |
| 5 | Dead |

<sup>\*</sup> As published in Am. J. Clin. Oncol.:

Oken, M.M., Creech, R.H., Tormey, D.C., Horton, J., Davis, T.E., McFadden, E.T., Carbone, P.P.: Toxicity And Response Criteria Of The Eastern Cooperative Oncology Group. Am J Clin Oncol 5:649-655, 1982.


# 10.6 Appendix: Protocol Amendment History

### 10.6.1 Amendment 1: 11 November 2021

#### **Overall Rationale for the Amendment:**

Protocol was moved to a new template allowing clarifications and further instruction to the study design to be made.

# Summary change table from previous version of the protocol

Any new or amended text in the protocol is indicated in bold. Deletions are marked in strikeout text. Minor formatting and editing are not included.

| Section | Was (Version1.0, 31 July 2019) | | Is (Version 2.0, 1 | 1 November 2021) | Rationale |
|---|---|---|---|---|---|
| Throughout | | | | te. Not all changes are identified. changes that impact the conduct in the amendment form. | New protocol template implemented |
| Throughout | Subject(s) | | Participant(s) | | New template<br>terminology |
| 1.1 / Synopsis<br>(Objectives/<br>Endpoints)<br>&<br>3 / Objectives and<br>Endpoints | Primary Objective(s) • To evaluate the efficacy of triptorelin pamoate 22.5 mg 6-month formulation in achieving castrate levels of testosterone (<50 ng/dL or <1.735 nmol/L) on Day 29 (i.e. 28 days after study drug injection) • Percentage of participants achievals of castrate levels of serum testosteron (<50 ng/dL or 1 nmol/L) on Day (i.e. 28 days after study drug injection) | eving<br>ne<br>735<br>29 | Primary Objectives(s) • To evaluate the efficacy of triptorelin pamoate 22.5 mg 6-month formulation in achieving castrate levels of testosterone | Primary Endpoint(s) Percentage of participants achieving castrate levels of serum testosterone (<50 ng/dL or 1.735 nmol/L) on Day 29 | Objectives and endpoint presentation made consistent with new protocol template guidance |


| Section | Was (Version1.0, 31 July 2019) | | Is (Version 2.0, 11 | November 2021) | Rationale |
|---|---|---|---|---|---|
| | To evaluate the efficacy of triptorelin pamoate 22.5 mg 6-month formulation in maintaining the castrate levels of serum testosterone from Week 8 to end of Week 24 in participants with locally advanced or metastatic prostate enneer | Percentage of<br>participants<br>maintaining the<br>castrate levels from<br>Week 8 to Week 24 in<br>participants with<br>locally advanced or<br>metastatic prostate<br>cancer | To evaluate the efficacy of triptorelin pamoate 22.5 mg 6-month formulation in maintaining the castrate levels of serum testosterone | Percentage of participants<br>maintaining the castrate<br>levels from Week 8 to<br>Week 24 | |

| D A | | | 100 |
|-----|----|-----|-----|
| -A | GE | 0// | 92 |

| Section | Was (Version1. | 0, 31 July 2019) | Is (Version 2.0, 11 | l November 2021) | Rationale |
|---|---|---|---|---|---|
| 1.1 / Synopsis (Objectives/ Endpoints) & 3 / Objectives and Endpoints | Secondary Objective(s) • To assess the safety of triptorelin pamoate 22.5 mg 6-month formulation over the study treatment period, i.e. from treatment start to 24 weeks | Secondary Endpoint(s) • Adverse events • Physical examination, ECG and vital signs • Laboratory parameters (haematology and blood chemistry) | Secondary Objective(s) • To assess the safety profile including local tolerability of triptorelin pamoate 22.5 mg 6-month formulation | Secondary Endpoint(s) Incidence of TEAEs (including local tolerability) throughout the study, i.e up to Week 24 Change from baseline in clinical safety laboratory parameters (blood chemistry and haematology) at Week 24 Change from baseline in physical examination at Day 1, Week 12 and Week 24 Change from baseline in ECG at Week 4 and Week 24 Change from baseline in vital signs (blood pressure and heart rate) at each visit up to Week 24 | Objectives and endpoint presentation made consistent with new protocol template guidance |

| PAGE 68/92 | 68/92 | GE | ${f PA}$ |
|------------|-------|----|----------|
|------------|-------|----|----------|

| Section | Was (Version1. | 0, 31 July 2019) | | Is (Version 2.0, 1 | l November 2021) | Rationale |
|---|---|---|---|---|---|---|
| | Primary Objective(s) | Primary Endpoint(s) | Τ | Secondary Objective(s) | Secondary Endpoint(s) | |
| | To assess the change in prostate specific antigen (PSA) levels from baseline throughout treatment | Change in PSA from<br>baseline (prior to<br>injection) on Week 12<br>and Week 24 | | To demonstrate the effect<br>of triptorelin pamoate<br>22.5 mg 6-month<br>formulation on PSA<br>response | Percent change in PSA from baseline (prior to injection) at Week 12 and Week 24 (Percent change in PSA is defined as the absolute value of difference between the PSA values at Week 12 and Week 24 and the baseline value divided by the baseline value) | |


| Section | Was (Version1.0, 31 July 20 | 019) | Is (Version 2.0, 1 | 1 November 2021) | Rationale |
|---|---|---|---|---|---|
| 1.1 / Synopsis (Objectives/ Endpoints) & 3 / Objectives and Endpoints | Secondary Pharmacokinetic/Phar | in PK<br>rs:-t <sub>max</sub> , C <sub>max</sub> ,<br>and AUC <sub>last</sub> | Secondary Objective(s) To assess the PK of triptorelin pamoate 22.5 mg 6-month formulation in a subset of 12 participants To assess the PD of testosterone in a subset of 12 participants To assess the PK of triptorelin pamoate 22.5 mg 6-month formulation for all participants To assess the PD of testosterone for all participants Exploratory To evaluate the PK/PD relations | Secondary Endpoint(s) PK parameters for dosing interval up to 24 weeks: otmax oCmax oAUC0-169 oAUClast PD parameters for dosing interval up to 24 weeks otmax oCmax otcast Sparse plasma concentrations of triptorelin at pre-dose and at Weeks 4, 8, 12, 16, 20 and 24 Sparse serum concentrations of testosterone at pre-dose and at Weeks 4, 8, 12, 16, 20 and 24 | Objectives and endpoint presentation made consistent with new protocol template guidance |


|---|---|---|---|
| 1.1 / Synopsis<br>(Sample Size<br>Determination) | Sample size is calculated to fulfil the co-primary efficacy criteria of this study, which is to assess the proportion of subjects achieving castrate levels of testosterone on Day 29 and the proportion of subjects maintaining the castrate levels of serum testosterone from Week 8 to end of Week 24. A total of 195 subjects with advanced prostate cancer will be enrolled to receive the triptorelin pamoate 22.5 mg 6 month formulation. [] Assuming the dropout rate will be around 15%, a sample size of 195 subjects in total is planned for this study. | Sample size is calculated to fulfil the co-primary efficacy criteria of this study, which is to assess the proportion of participants achieving castrate levels of testosterone on Day 29 and the proportion of participants maintaining the castrate levels of serum testosterone from Week 8 to end of Week 24. [] Assuming the dropout rate will be around 15%, a sample size of 195 participants with locally advanced or metastatic prostate cancer in total is planned for this study. | Removal of repetition in the text |
| 1.1 / Synopsis<br>(Primary Analysis)<br>&<br>9.4.2 / Analysis of<br>Primary Endpoints | The proportion of subjects who achieved castration levels of serum testosterone on Day 29 and the proportion of subjects who maintained the levels from Week 8 to end of Week 24 will be tabulated with two-sided 95% confidence interval (95% CI) using the binomial distribution. | Co-primary endpoints will be tabulated with two-sided 95% confidence interval (95% CI) using the Clopper-Pearson exact method. | Removal of repetition in<br>the synopsis and<br>clarification of analysis |

D-CN-52014-237

|---|---|---|---|
| 1.3 / Schedule of<br>Activities | The schedule of activities during the study is summarised for all subjects, except the PK/PD subset of subjects in Table 1 and for the PK/PD subset of participants in Table 2. | The schedule of activities during the study is summarised for all participants in Table 1, except the PK/PD subset of 12 participants which is summarised in Table 2. If the COVID-19 pandemic prevents participants from coming to the site, participants can have their study visit assessments performed remotely as judged appropriate by the investigator. This must be discussed with the sponsor before being implemented. In such a case, the investigator will perform a telemedicine visit and will make every effort, where applicable, to contact the participant's general practitioner or specialist physician to ensure all important medical information and safety event(s) occurring since the last visit are collected. Guidance on how to collect protocolplanned assessments will be provided to the investigator in a separate document. Such document will be filed in the trial master file. Independent ethics committees (IECs)/institutional review boards (IRBs) will be notified of the changes as applicable locally. Of note, as the adapted | Guidance for COVID-19 management during the study added per new template. |
| 1.3 / Schedule of<br>Assessments | | visit deviates from the regular protocol plan, the changes will be recorded as protocol deviations related to COVID-19. The following assessments were added for screening in Table 1 and Table 2: Demography MRI scan [g] for Table 1 [h] for Table 2 Footnote "g" and "h": Scan for prostate gland or the whole body, only if necessary, based on investigator's judgement. An MRI scan is not required if performed within 1 month of screening. | Clarification of procedures required at screening |
| 1.3 / Schedule of<br>Assessments<br>(Table 1 and<br>Table 2) | Medical history | Medical and surgical history | Clarification of information to be collected at screening |


| G | W (V11 0 21 T-12010) | | | T- (V | | D // 1 | |
|---|---|---|---|---|---|---|---|
| 1.3 / Schedule of<br>Assessments<br>(Table 1 and<br>Table 2) | Physical examination | | [g<br>C<br>P<br>a | hysical examination [f] for Table 1 g] for Table 2 corresponding footnote "f" and "g": articipants, particularly those wit dvised regarding clinical signs succession. | | | |
| 1.3 / Schedule of | Disease history and previous | x | | Disease-specific medical history | | X | Clarification of collection |
| Assessments | treatment | Λ | | Prior disease-specific treatment | , | X | of prior treatments as |
| (Table 1 and<br>Table 2) | | | | - | | | screening for prostate<br>cancer |
| 1.3 / Schedule of | Blood sample for | X X | | Blood sample for testosterone | X | X [a, | Clarification added to |
| Assessments<br>(Table 1 and | testosterone PD | [e] | | PD | | e] | footnote "a" that sampling should occur pre-dose on |
| Table 2) | | | | | | | Day 1 |
| 1.3 / Schedule of | Blood sample [c] for | X X | | Blood sample [c] for | X | X [a, | Clarification of |
| Assessments<br>(Table 1) | laboratory safety tests | [e] | | laboratory safety tests | | e] | assessment timing on<br>Day 1 |
| 1.3 / Schedule of<br>Assessments | Blood sample [d] for laboratory safety tests | X X [f] | + | Blood sample [c] for laboratory safety tests | X | X [a, | Clarification of assessment timing on |
| (Table 2) | laboratory sarety tests | | | laboratory safety tests | | 1 1 | Day 1 |
| 1.3 / Schedule of<br>Assessments<br>(Table 2) | Blood sample for triptorelin PK | X X [c] | | Blood sample for triptorelin<br>PK | X | X [a,<br>c] | Clarification of<br>assessment timing on<br>Day 1 |
|---|---|---|---|
| 1.3 / Schedule of<br>Assessments<br>(Table 1 and Table<br>2) | Blood samples for PSA | Blood samples for PSA X | PSA added at screening<br>for consistency with<br>eligibility requirements |
| 1.3 / Schedule of<br>Assessments<br>(Table 1 and Table<br>2) | Previous and concomitant medication | Previous (excluding disease-specific) and concomitant medication | Clarification that other<br>prior medication<br>collection excludes<br>disease-specific<br>treatments |
| 1.3 / Schedule of<br>Assessments<br>(Table 1 and Table<br>2) | Footnote "c" Haematology (WBC, Platelet count, Hb), Blood Chemistry (creatinine, glucose, ALT, AST, alkaline phosphatase, bilirubin). Glucose: Non-fasting levels in all participants at Screening visit, fasting levels on Days 1 and 169. Fasting is not necessary for diabetic participants. | Footnote "c" Haematology (WBC, platelet count, Hb), Blood Chemistry (creatinine, glucose, ALT, AST, alkaline phosphatase, bilirubin (total and conjugated)). Glucose: Fasting levels in all participants at Screening visit, fasting levels on Days 1 and 169. Fasting is not necessary for diabetic participants. | Clarification of bilirubin<br>and glucose collection |
| 2.1 / Study<br>Rationale | At the same time, triptorelin pharmacokinetics (PK) and testosterone pharmacodynamics (PD) will be assessed in a subset of 12 Chinese subjects. | In addition, triptorelin pharmacokinetics (PK) and testosterone pharmacodynamics (PD) will be assessed in the study population. | Clarification of study<br>procedures |
| 2.2 / Background | Further details/additional information regarding risks and benefits to human subjects may be found in the Investigator's Brochure. | | Removal of repetition<br>with other sections in the<br>protocol |
| 2.3 / Benefit/Risk<br>Assessment | | Detailed information about the known and expected benefits and risks and reasonably expected adverse events (AEs) of triptorelin may be found in the IB. | Addition per new template |

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024


| 2.3.1 / Risk<br>Assessment | A risk assessment for this study is provided in Table 3. Table 3 Study Risk Assessment Addition per new template |
|---|---|
| | Potential Risk of Clinical Significance Summary of Data/Rationale for Risk Mitigation Strategy |
| | Study Intervention: Triptorelin |
| | There is no major known nonclinical risk associated with the study intervention Clinical risks associated with the study intervention may include: • hot flushes • erectile dysfunction • loss of libido • impaired physical activities • metabolic syndrome • cardiovascular events • anxiety/depression • decreased bone mineral density • risk of abortion or foetal abnormality [b] |
| | See Section 8.3 including local tolerability |


| Section | Was (Version1.0, 31 July 2019) | Is (Version 2.0 | ), 11 November 20 | )21) | Rationale |
|---|---|---|---|---|---|
| | | There are no specific risks related to the study design or procedures. IB=investigator's brochu | | | |
| | | a Pregnancy is not releve<br>However, reproductive r | | | |
| | | for female partners of pa | | | |
| | | pregnant. | тастранто ино ша | iy become | |

|------------|
|------------|

|---|---|---|---|
| 2.3.2 / Benefit<br>Assessment | | Based on the nonclinical and clinical data generated up to finalisation of the protocol, treatment with triptorelin 6-month formulation may maintain castrate levels of testosterone for a longer period i.e. 6 months (24 weeks), thereby reducing the need for frequent injections, in Chinese participants with locally advanced or metastatic prostate cancer to a similar extent as in a previous global phase III study. | Addition per new template |
| 2.3.3 / Overall<br>Benefit: Risk<br>Conclusion | | Taking into account the measures taken to minimise risk to participants, the potential risks identified in association with triptorelin are justified by the anticipated benefits that may be afforded to Chinese participants with locally advanced or metastatic prostate cancer. | Addition per new template |
| 4.3 / Justification<br>for Dose | | For this intervention, the term "dose" refers to the i.m. injection of triptorelin 22.5 mg created to guarantee the release of a monthly dose of 3.75 mg over a 169-day period. In addition, results from a phase III study have shown the 6-month triptorelin 22.5 mg formulation to induce and maintain castration in participants with locally advanced or metastatic prostate cancer, as well as demonstrate a good safety profile [Lundstrom 2009]. | Addition per new template |
| 4.4 / End of Study<br>Definition | This study will consist of a 4-week screening period, a single open-label administration of the IMP on Day 1 followed by an assessment period of 24 weeks. Subjects are expected to participate in this study for the entire 24 weeks. The subject's participation in the study will be considered to have ended at the time of the last visit. The overall duration of the study (from first subject in to last subject out) will be approximately 30 months. The study will be considered to have started when the first subject has provided signed informed consent. | The end of the study (EoS) is defined as the date of the last visit of the last participant in the study as shown in the SoA (Table 1 and Table 2). The overall duration of the study (from first participant in, to last participant out) will be approximately 30 months. The study will be considered to have ended after the last participant has completed the last visit (at Week 24) in the study. A participant is considered to have completed the study if they have completed all phases of the study including the last visit. Criteria for study intervention discontinuation and participant discontinuation/withdrawal from the study are described in Section 7.1 and Section 7.2, respectively. Loss to follow-up is described in Section 7.3. | Updated per new template |

|---|---|---|---|
| | The study will be considered to have ended after the last subject has completed the last follow up period (at Week 24) in the study. | | |
| 5.1 / Inclusion<br>Criteria | Signed written informed consent before entry into the study. A histologically or cytologically confirmed, locally advanced or metastatic prostate cancer, and should be staged T3-4NxM0 or TxN1M0 or TxNxM1 according to the TNM classification or participant should have rising PSA after failed local therapy and be a candidate for androgen deprivation therapy (ADT). | 1. Participant is capable of giving signed informed consent as described in Appendix 10.1 which included compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. 3. Has a histologically or cytologically confirmed adenocarcinoma, locally advanced or metastatic prostate cancer which is staged T₃₄NxM0 or TxN1M0 or TxNxM1 according to the TNM classification. Or participant has PSA recurrence after curative treatment and be a candidate for androgen deprivation therapy (ADT). (Note: PSA recurrence after radical prostatectomy: PSA ≥0.2 ng/mL and rising, confirmed on a repeat test; PSA recurrence after radiation therapy: PSA increased 2 ng/mL than the lowest level.) 8. Participant is male 9. Male participants must agree that, if their partner is at risk of becoming pregnant, they will use an effective method of contraception. The participant must agree to use the contraception during the whole period of the study and for 9 months after the last dose of study intervention. | Addition per new template |
| 5.2 / Exclusion<br>Criteria | | 4. Metastatic hormone-sensitive prostate cancer with high tumour burden | Clarification of participant eligibility |
| 5.2 / Exclusion<br>Criteria | 19. Inability to give informed consent or to comply fully with the protocol. | | Removal of duplication<br>with inclusion #1 |


|---|---|---|---|
| 5.3 / Lifestyle<br>Considerations | | Participants will be advised to avoid chronic alcohol use and smoking during the study. | Addition per new template |
| 5.4 / Screen<br>Failures | Under no circumstances will subjects be screened more than once. | A screen failure occurs when a participant who consents to participate in the clinical study is not subsequently entered in the study. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants to meet the Consolidated Standards of Reporting Trials (CONSORT) publishing requirements and to respond to queries from regulatory authorities. Minimal information includes date of informed consent, demography, reason for screen failure, eligibility criteria and any serious adverse event (SAE). Individuals who do not meet the criteria for participation in this study (screen failure) will not be rescreened. | Addition and clarification per new template |
| 6.8 / Concomitant<br>Therapy | | Any medication (excluding prior disease-specific medications) or vaccine (including over the counter prescription medicines, recreational drugs, vitamins, and/or herbal supplements) that the participant had received within 2 months before triptorelin administration or during triptorelin administration must be recorded on the eCRF along with: [] | Addition per new<br>template and clarification<br>that prior medications<br>exclude those for previous<br>disease-specific treatment |
| 6.8 / Concomitant<br>Therapy | Any treatment or procedure with an effect on androgenic hormones be administered concomitantly to the study drug (will be considered as a protocol violation). | <ul> <li>Any treatment or procedure with a specific or potential effect on androgenic hormones be administered concomitantly to the study drug (will be considered as a protocol violation). Per investigator's clinical judgement, suggest offering short-term administration of an older generation androgen receptor antagonist to M1 participants starting study intervention to reduce the risk of the 'flare-up' phenomenon.</li> <li>Any medication which raises prolactin levels and those affecting pituitary secretion of gonadotropins</li> </ul> | Clarification of medications not permitted during the study |


#### PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024

|---|---|---|---|
| 6.8 / Concomitant<br>Therapy | [] • Other medications: any treatment including analgesics, which is considered necessary for the participant's welfare, may be given at the discretion of the investigator | <ul> <li>Anticonvulsants (e.g phenobarbital): long-term therapy may have additional risk for osteoporosis.</li> <li>Other medications: any treatment which is considered necessary for the participant's welfare, may be given at the discretion of the investigator.</li> </ul> | Clarification of<br>medication use that<br>should be monitored<br>during the study |
| 7.1 /<br>Discontinuation of<br>Study Intervention | | In this study, there will only be one treatment cycle administered on Day 1 of the study, thus discontinuation of the study intervention is not applicable (i.e. no repeat cycles). In the event a participant is enrolled, but does not receive study intervention, the participant will not remain in the study and EoS/EW assessment will not be performed. Only the reason for discontinuation will be collected. | Addition per new template |
| | | If participants are lost to follow-up, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law. | |
| 7.1.1 / Temporary<br>Discontinuation | | In case of suspected or confirmed COVID-19 (SARS-CoV-2) infection, the intervention administration may be temporarily postponed depending on the participant clinical presentation. In some cases, the investigator may request a participant be retested before the intervention administration. | Guidance for COVID-19<br>management during the<br>study added per new<br>template. |


|---|---|---|
| 7.3 / Lost to<br>Follow-up | A participant will be considered lost to follow-up if they repeatedly fail to return for scheduled visits and is unable to be contacted by the study site. | Addition per new template |
| | The following actions must be taken if a participant fails to return to the clinic for a required study visit: | |
| | <ul> <li>The site must attempt to contact the participant and<br/>reschedule the missed visit as soon as possible. The<br/>site should counsel the participant on the importance<br/>of maintaining the assigned visit schedule and<br/>ascertain whether the participant wishes to and/or<br/>should continue in the study.</li> </ul> | |
| | Before a participant is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the participant (where possible, three telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods). These contact attempts should be documented in the participant's medical record. | |
| | <ul> <li>Should the participant continue to be unreachable,<br/>he/she will be considered to have withdrawn from the<br/>study.</li> </ul> | |
| | Site personnel will attempt to collect the vital status of the participant within legal and ethical boundaries for all participants enrolled, including those who did not receive study intervention. Public sources may be searched for vital status information. If vital status is determined as deceased, this will be documented, and the participant will not be considered lost to follow-up. Sponsor personnel will not be involved in any attempts to collect vital status information. | |
| 8.1 / Demography | Age, sex and, according to individual country regulations/requirements and if authorised in the country, ethnicity will be collected. | Addition per new template |


| PROTOCOL | · FINAL with | Amendment 3: Version 4.0. 08 | March 2024 |
|----------|--------------|------------------------------|------------|

|---|---|---|---|
| 8.2 / Efficacy<br>Assessments | | Approximately 26 mL of blood will be collected from all participants, and approximately 38 mL of blood from the PK/PD subset participants, for measurement of testosterone and PSA. Serum samples used to evaluate testosterone and PSA will be divided into two aliquots (one primary and one back-up). Further instructions for the collection, handling and shipment of biological samples will be provided by the | Clarification of efficacy<br>assessments and blood<br>collection |
| 8.2.1 /<br>Testosterone | Testosterone will be assessed by a third-party vendor, as described in the Laboratory Manual according to the analytical procedure described above in Section 9.1.2. | Testosterone will be assessed by a third-party vendor, as described in the Laboratory Manual. Serum will be analysed to determine concentrations of testosterone using a validated, specific and sensitive liquid chromatography tandem mass spectrometry (LC-MS/MS) methods. [] Residual serum samples remining from the analysis may also be retained by the sponsor for additional investigations. This could include using leftover serum for long-term stability, reproducibility, or other bioanalytical assessments. Surplus serum samples may be used in China or shipped outside China as required. Surplus serum samples will be managed anonymously and will not be identifiable. | Clarification of efficacy assessment method. |
| 8.3.1 / Physical<br>Examination | | In addition, participants, particularly those with M1b status, should be advised regarding clinical signs suggestive of spinal cord compression. | Clarification of procedures for physical examination |
| 8.3.2 / Vital Signs | Blood pressure and heart rate will be assessed at timepoints described in Table 1 with an automated device so that measurements are independent of the observer. | Blood pressure, temperature, respiratory rate and heart rate will be assessed as outlined in the SoA (Section 1.3) with an automated device so that measurements are independent of the observer. Any clinically significant vital signs will be recorded as AEs. | Clarification of collection of vital sign data |


|---|---|---|---|
| 8.3.3 /<br>Electrocardiograms | Twelve lead ECGs will be recorded so that the different ECG intervals (RR, PR, QRS, QT, QTcF) can be measured automatically. | A single 12-lead ECG will be recorded so that the different ECG intervals (RR, PR, QRS, QT, QTcF) can be measured automatically. | Clarification of data collection |
| 8.3.4 / Magnetic<br>Resonance<br>Imaging Scan | | 8.3.4 Magnetic Resonance Imaging Scan A magnetic resonance imaging scan for prostate gland or whole body (only if necessary, based on investigator's judgement) will be performed as described in the SoA (Table 1 and Table 2) to confirm disease stage prior to study entry. An MRI scan is not required, if performed within 1 month of study screening. | Additional procedures at screening |
| 8.3.6 / Local<br>Tolerance | Local tolerance will be assessed at 2 and 4 hours after injection. | Local tolerance will be assessed 2 hours after injection. | Simplified to improve participant compliance with study procedures |
| 8.4.8 / Reporting<br>of Study<br>Intervention Errors<br>Including<br>Misuse/Abuse | | <ul> <li>Medication errors are unintentional errors in the<br/>prescribing, storing, dispensing, preparing or<br/>administration of a study intervention (medicinal<br/>product) while under the control of a healthcare<br/>professional, participant or consumer.</li> </ul> | Added per new template |
| | | <ul> <li>Misuse refers to situations where the study<br/>intervention is intentionally and inappropriately<br/>used not in accordance with the protocol.</li> </ul> | |
| | | <ul> <li>Abuse corresponds to the persistent or sporadic,<br/>intentional excessive use of a medicinal product,<br/>which is accompanied by harmful physical or<br/>psychological effects.</li> </ul> | |
| | | <ul> <li>Study intervention errors and uses outside of what is foreseen in the protocol will be recorded in the eCRF irrespective of whether associated with an AE/SAE or not. It will also be documented in the AE section of the eCRF if associated with an AE. It will be reported in the safety database only if associated with an SAE.</li> </ul> | |

| D A | | 02 | 100 |
|------------------|------------|----|-----|
| $\mathbf{P}_{P}$ | <b>LGE</b> | 03 | 92 |

|---|---|---|---|
| 9.1 / Statistical<br>Hypothesis | | No statistical hypotheses are planned for this study. | Addition per new template |
| 9.4 / Statistical<br>Analysis | | The statistical analysis plan (SAP) will be finalised before the first participant enters the study and it will include a more technical and detailed description of the statistical analyses described in this section. This section is a summary of the planned statistical analyses of the most important endpoints including primary and key secondary endpoints. | Addition per new template |
| | | Other endpoints as well as demographic, baseline characteristics and disposition will be detailed in the SAP. | |
| | | Statistical evaluation will be performed using Statistical Analysis System (SAS®) Version 9.4 (or higher if available). | |
| 9.4.2 / Analysis of | The co-primary efficacy variables are | The co-primary efficacy variables are | Endpoint presentation<br>made consistent with new<br>protocol template<br>guidance |
| Primary Endpoints | • percentage of participants achieving castrate levels of<br>serum testosterone (<50 ng/dL or 1.735 nmol/L) 4 | • percentage of participants achieving castrate levels of serum testosterone (<50 ng/dL or 1.735 nmol/L) and | |
| | weeks after the first injection and • percentage of participants maintaining the castrate levels from Week 8 to Week 24 in participants with locally advanced or metastatic prostate cancer. | • percentage of participants maintaining the castrate levels from Week 8 to Week 24. | gurdanee |
| 9.4.3.1 / Prostate-<br>specific Antigen | The secondary efficacy variable is the change in PSA from baseline (prior to injection) measured at Week 12 and Week 24. | The secondary efficacy variable is the percent change in PSA from baseline (prior to injection) measured at Week 12 and Week 24. Percent change in PSA is defined as the absolute value of difference between the PSA values at Week 12 and | Endpoint presentation<br>made consistent with new<br>protocol template<br>guidance |
| | The efficacy analysis will be presented for the FAS and PP population. The main analysis will be conducted in the FAS population. | Week 24 and the baseline value divided by the baseline value. The efficacy analysis for the primary and secondary efficacy endpoints will be presented for the FAS and PP population. The analysis of the safety data will be performed based on the safety set and analysis of PK and PD in the relevant PK analysis set. | |

| GE. |
|-----|

|---|---|---|---|
| 9.4.3.2 / Pharmacokinetic and Pharmacodynamic Data Analysis | | [] Individual and mean triptorelin and testosterone concentration time profiles, as well as spaghetti plots, will be generated. | Clarification of planned analysis |
| 9.4.3.2 /<br>Pharmacokinetic<br>and<br>Pharmacodynamic<br>Data Analysis | Non-compartmental Analysis The PK analysis of triptorelin plasma concentrations and testosterone serum concentrations of the rich sampling PK/PD subgroup will be performed by NCA approach using Phoenix WinNonlin PK program version 6.3 or higher. | Non-compartmental Analysis The PK analysis of triptorelin plasma concentrations and testosterone serum concentrations of the rich sampling PK/PD subset will be performed by NCA approach using Phoenix WinNonlin PK program version 8.3 or higher. | Clarification of planned analysis |
| 9.4.3.2 / Pharmacokinetic and Pharmacodynamic Data Analysis | Population Pharmacokinetic Analysis Population pharmacokinetics (PopPK) modelling will be performed to characterise triptorelin PK parameters, such as (but not restricted to) clearance (apparent total clearance, CL/F) and volume of distribution (apparent volume of distribution, V/F), as well as their interindividual variability. | Population Pharmacokinetic Analysis Population pharmacokinetics (PopPK) modelling will be performed using concentrations obtained from all participants in order to describe the pharmacokinetics of triptorelin 6-month formulation in the prostate cancer population (if warranted by the data). In addition, quantification of the inter-participant variability on PK will be performed and an attempt to identify participant characteristics explaining the variability on PK will be made. The PK model developed will be used to derive exposure metrics to perform an exploratory analysis with efficacy and safety endpoints (should any safety signal emerge). Should a trend be observed, PK/PD modelling will be performed to describe the relationship between exposure and efficacy and/or safety endpoints. Population PK/PD analysis will be described in a separate data analysis plan and presented in a stand-alone report. | Clarification of planned analysis |


#### 10.6.2 Amendment 2: 07 April 2022

#### **Overall Rationale for the Amendment:**

Protocol was updated to clarify definition of primary endpoints and change safety laboratory testing from central to local during the study.

#### Summary change table from previous version of the protocol

Any new or amended text in the protocol is indicated in bold. Deletions are marked in strikeout text. Minor formatting and editing are not included.

| Section | Was (Version 2.0, 11 I | lovembei | r 2021) | Is (Version 3.0, 07 | April 2 | 2022) | Rationale |
|---|---|---|---|---|---|---|---|
| 1.3 / Schedule of<br>Activities<br>(Table 1) | Blood sample for<br>testosterone PD<br>Blood samples for PSA | X | X [a, e]<br>X [a] | Blood sample for<br>testosterone PD [h]<br>Blood samples for<br>PSA [h] | X | X [a, e] | Clarification of laboratory testing location. |


| Section | Was (Version 2.0, 11 November 2021) | Is (Version 3.0, 07 April 2022) | Rationale |
|---|---|---|---|
| 1.3 / Schedule of Activities (Table 1 Footnotes) | c Haematology (WBC, platelet count, Hb), Blood Chemistry (creatinine, glucose, ALT, AST, alkaline phosphatase, bilirubin (total and conjugated)). Glucose: fasting levels in all participants at Screening visit, fasting levels on Days 1 and 169. Fasting is not necessary for diabetic participants. d Injection site to be specifically checked 2 and 4 hours after injection for local reactions on Day 1. After Day 1, any local reaction AE to be collected on the CRF in the same manner as other AEs. e Measurement of testosterone and laboratory safety tests for analysis purposes only and not for eligibility—the screening testosterone and safety laboratory test results will be used for eligibility. f Participants, particularly those with M1b status, should be advised regarding clinical signs suggestive of spinal cord compression. | c Haematology (WBC, platelet count, Hb), Blood Chemistry (creatinine, glucose, ALT, AST, alkaline phosphatase, bilirubin (total and conjugated)) will be tested at the local laboratory. Glucose: fasting levels in all participants at Screening visit, fasting levels on Days 1 and 169. Fasting is not necessary for diabetic participants. d Injection site to be specifically checked 2 hours after injection for local reactions on Day 1. After Day 1, any local reaction AE to be collected on the CRF in the same manner as other AEs. e Measurement of testosterone, PSA and laboratory safety tests for analysis purposes only and not for eligibility. The screening testosterone, PSA and safety laboratory test results will be used for eligibility. f Complete physical examination to be performed (or brief physical examination based on investigator judgement). Participants, particularly those with M1b status, should be advised regarding clinical signs suggestive of spinal cord compression. h Testosterone and PSA testing will be performed at the central laboratory. | Clarification of laboratory testing location and study procedures. |
| 1.3 / Schedule of<br>Activities | Blood sample for triptorelin PK X [a, c] | Blood sample for triptorelin PK X [c] | Removed reference to footnote "a" to avoid confusion with footnote "c". |
| (Table 2) | Blood sample for testosterone PD X X [a, f] | Blood sample for testosterone PD [i] X X [a, f] | Clarification of laboratory testing location. |
| | Blood sample for PSA X X [a] | Blood sample for PSA X X [a, f] | |


| PROTOCOL | FINAL wi | ith Amendmen | t 3: Version | 4 0 0 | 8 March 2024 |
|----------|----------|--------------|--------------|-------|--------------|

| Section | Was (Version 2.0, 11 November 2021) | Is (Version 3.0, 07 April 2022) | Rationale |
|---|---|---|---|
| 1.3 / Schedule of | d Haematology (WBC, platelet count, Hb), Blood | d Haematology (WBC, platelet count, Hb), | Clarification of laboratory testing location |
| Activities | Chemistry (creatinine, glucose, ALT, AST, alkaline | Blood Chemistry (creatinine, glucose, ALT, | and study procedures. |
| (Table 2 | phosphatase, bilirubin (total and conjugated). | AST, alkaline phosphatase, bilirubin (total and | |
| Footnotes) | Glucose: Fasting levels in all participants at | conjugated) will be tested at the local | |
| | Screening visit, fasting levels on Days 1 and 169. | laboratory. Glucose: Fasting levels in all | |
| | Fasting is not necessary for diabetic participants. | participants at Screening visit, fasting levels on | |
| | | Days 1 and 169. Fasting is not necessary for | |
| | e Injection site to be specifically checked 2 <del>and 4</del> | diabetic participants. | |
| | hours after injection for local reactions on Day 1. | | |
| | After Day 1, any local reaction AE to be collected on | e Injection site to be specifically checked | |
| | the CRF in the same manner as other AEs. | 2 hours after injection for local reactions on | |
| | | Day 1. After Day 1, any local reaction AE to be | |
| | f Measurement of testosterone and laboratory safety | collected on the CRF in the same manner as | |
| | tests for analysis purposes only and not for eligibility | other AEs. | |
| | —the screening testosterone and safety laboratory | | |
| | test results will be used for eligibility. | f Measurement of testosterone, PSA and | |
| | | laboratory safety tests for analysis purposes | |
| | g Participants, particularly those with M1b status, | only and not for eligibility. The screening | |
| | should be advised regarding clinical signs suggestive | testosterone, PSA and safety laboratory test | |
| | of spinal cord compression. | results will be used for eligibility. | |
| | | g Complete physical examination to be | |
| | | performed (or brief physical examination | |
| | | based on investigator judgement). | |
| | | Participants, particularly those with M1b status, | |
| | | should be advised regarding clinical signs | |
| | | suggestive of spinal cord compression. | |
| | | i Testosterone and PSA testing will be | |
| | | performed at the central laboratory. | |


| Section | Was (Version 2.0, 11 November 2021) | Is (Version 3.0, 07 April 2022) | Rationale |
|---|---|---|---|
| 7.2 / Participant Discontinuation/ Withdrawal from the Study | A participant may withdraw from the study at any time at his/her own request or may be withdrawn at any time at the discretion of the investigator for safety, behavioural or compliance reasons. A participant may be withdrawn from the study for any of the following reasons including: O Drug related AE O Non drug related AE O Participant lost to follow-up O Non drug related reason, e.g. the participant relocates At the time of discontinuing from the study, if possible, an early discontinuation visit should be conducted, as shown in the SoA. See SoA for data to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed. | <ul> <li>A participant may withdraw from the study at any time at his/her own request or may be withdrawn at any time at the discretion of the investigator for safety, behavioural or compliance reasons.</li> <li>At the time of discontinuing from the study, an early discontinuation visit should be conducted, as shown in the SoA. See SoA for data to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed.</li> </ul> | Removed for conciseness as reasons for withdrawal will be presented in the electronic case report form. |
| 8.1 / Demography | Age, sex and, according to individual country regulations/requirements and if authorised in the country, ethnicity will be collected. | Age, sex and, according to individual country regulations/requirements and if authorised in the country, race/ethnicity will be collected. | Clarification of demographic information to be collected. |
| 8.2.1 /<br>Testosterone | Residual serum samples remining from the analysis may also be retained by the sponsor for additional investigations. This could include using leftover serum for long-term stability, reproducibility, or other bioanalytical assessments. Surplus serum samples may be used in China or shipped outside China as required. Surplus serum samples will be managed anonymously and will not be identifiable. | Residual serum samples remining from the analysis may also be retained by the sponsor for <b>up to 5 years after completion of the study</b> . This could include using leftover serum for long-term stability <b>or</b> reproducibility assessments. Surplus serum samples <b>can only</b> be used in China. Surplus serum samples will be managed anonymously and will not be identifiable. | Clarification of sample use. |

| Section | Was (Version 2.0, 11 November 2021) | Is (Version 3.0, 07 April 2022) | Rationale |
|---|---|---|---|
| 8.3.1 / Physical<br>Examinations | A complete physical examination will include, at a minimum, assessments of the cardiovascular, respiratory, gastrointestinal and neurological systems. Height and weight will also be measured and recorded. Body weight will be measured in underwear and without shoes. A brief physical examination will include, at a minimum, assessments of the skin, lungs, cardiovascular system, abdomen (liver and spleen). | A complete physical examination will include, at a minimum, assessments of the skin, and cardiovascular, respiratory, gastrointestinal and neurological systems. Height and weight will also be measured and recorded. Body weight will be measured in underwear and without shoes. A brief physical examination will include, at a minimum, assessments of the lungs, cardiovascular system, abdomen (liver and spleen). | Clarification of study procedures. |
| 8.3.5 / Clinical<br>Safety Laboratory<br>Assessments | •All clinical laboratory safety tests (haematology and blood biochemistry) will be assessed at a central laboratory (as described in the Laboratory Manual). Local testing can be performed optionally as required. | •All clinical laboratory safety tests (haematology and blood biochemistry) will be assessed locally. | To reduce complexity of obtaining safety assessments during study. |
| 8.5 /<br>Pharmacokinetics | <ul> <li>Surplus plasma samples may be used in China or shipped outside China; if required, for the purposes of eross validating the bioanalytical method/s used in this study. Surplus plasma samples will be managed anonymously and will not be identifiable.</li> <li>Residual plasma samples remaining from the analyses may also be retained by the sponsor for additional investigations. This could include using leftover plasma for long-term stability; reproducibility, or other bioanalytical assessments.</li> </ul> | <ul> <li>Surplus plasma samples will be used in China and will not be shipped outside China. Surplus plasma samples will be managed anonymously and will not be identifiable.</li> <li>Residual plasma samples remaining from the analyses may also be retained by the sponsor for up to 5 years after the completion of the study. This could include using leftover plasma for long-term stability or reproducibility assessments.</li> </ul> | Clarification of sample use. |
| 9.4.2 / Analysis of<br>the Primary<br>Endpoints | | The percentage of participants achieving castrate levels of serum testosterone (<50 ng/dL or 1.735 nmol/L) on Day 29 will be obtained as the number of participants with castrate levels at the visit, divided by the total number of participants on Day 29 in the considered population. | Clarification of definition for primary endpoints. |


| Section | Was (Version 2.0, 11 November 2021) | Is (Version 3.0, 07 April 2022) | Rationale |
|---|---|---|---|
| | | Percentage of participants maintaining the castrate levels of serum testosterone (<50 ng/dL or 1.735 nmol/L) from Week 8 to Week 24 will be calculated as the number of participants with castrate levels at all visits from Week 8 to Week 24, divided by the total number of assessable participants. | |
| | | To derive the percentage of participants maintaining castration levels of testosterone, missing data will be handled as follows: | |
| | | (a) In participants escaping castration at a certain visit, subsequent missing data is irrelevant. | |
| | | (b) Participants maintaining castration up to<br>a certain visit with missing data afterwards<br>(drop-out due to non-drug-related reasons)<br>will be excluded from the analysis. | |
| | | (c) Participants maintaining castration up to<br>a certain visit with missing data afterwards<br>(drop-out due to drug-related reasons) will be<br>treated as having escaped castration (failure). | |
| | | (d) Missing data between two visits where<br>castration levels are maintained will be<br>handled as missing for that particular visit,<br>and the participant will be considered to have<br>maintained castration. | |
| | | To derive the percentage of participants maintaining castrate levels of testosterone, assessable participants are defined as the total number of all participants having values at all visits and all participants having | |
| | | missing data according to the criteria a), c) and d) mentioned previously. Participants having missing data according to the criteria b) will be excluded from this calculation. | |


| Section | Was (Version 2.0, 11 November 2021) | Is (Version 3.0, 07 April 2022) | Rationale |
|---|---|---|---|
| 9.4.3.2 /<br>Pharmacokinetic<br>and<br>Pharmacodynamic<br>Data Analysis<br>(Population<br>Pharmacokinetic<br>Analysis) | | Historical PK data from other studies may also be used to compare the PK profiles from this study against other populations. | Clarification of potential pharmacokinetic analysis. |
| 10.1.8 / Study and<br>Site Start and<br>Closure | The study start date is the date on which the clinical study will be open for recruitment of participants. | The study start date is the date on which the clinical study will be open for recruitment of participants or the actual date on which the first participant is enrolled. | Statement made consistent with definition in 42 CFR 11.10(b) (16). |
| 10.2 / Appendix:<br>Clinical<br>Laboratory Tests | • The tests detailed in Table 6 will be performed by a central laboratory (local testing can be performed optionally as required). | • The tests detailed in Table 6 will be performed locally. | To reduce complexity of obtaining safety assessments during study. |
| 10.2 / Appendix:<br>Clinical<br>Laboratory Tests | Note: All parameters will be analysed eentrally. The preparation and storage of samples are described separately in the Laboratory Manual. Local tests will be conducted as optional extra tests as required by local sites. | Note: All parameters will be analysed locally. The preparation and storage of samples will be performed per each local laboratory practice. | To reduce complexity of obtaining safety assessments during study. |
| 10.3.2 / Definition<br>of SAEs | A suspected or confirmed coronavirus COVID-19 (SARS-CoV-2) infection must be reported as serious (seriousness criteria should be "other medically significant" if no other seriousness criteria are present (e.g. hospitalisation). | A suspected or confirmed coronavirus COVID-19 (SARS-CoV-2) infection should be reported as serious if the event meets the defined seriousness criteria. If no seriousness criteria are reported by the investigator, the COVID-19 event will be collected and recorded as nonserious. | Protocol template update. |

PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024 PAGE 92/92

#### 11 REFERENCES

Barron JL, Millar RP, Searle D: Metabolic clearance and plasma half-disappearance time of DTrp6 and exogenous luteinizing hormone-releasing hormone. J Clin Endocrinol Metab 1982; 54:1169-73.

Botto H et al.: Decapeptyl in the treatment of metastatic prostatic cancer. Comparative study with pulpectomy. Prog Biol Res 1987; 243A:199-206.

Breul J, Lundstrom EA, Purcea D et al. Efficacy of testosterone suppression with sustained-release triptorelin in advanced prostate cancer. Adv Ther. 2017;34(2):513-23.

De Sy WA, De Wilde P, De Meyer JM et al.: Long term experience in the treatment of advanced prostatic cancer with Decapeptyl, compared to orchiectomy. Acta Urol Belgica, 1988;56581-8.

Filicori M: Gonadotropin-Releasing Hormone Agonists - A guide to use and selection. Drugs 1994;48:41-58.

Huggins C, Hodges CV: Studies on prostatic cancer I. The effects of castration, of oestrogen, and of androgen injection on serum phosphatases in metastatic carcinoma of the prostate. Cancer Res 1941;1:293-7.

Huggins C, Stevens REJr, Hodges CV: Studies on prostate cancer II. The effects of castration on advanced carcinoma of the prostate gland. Arch Surg 1941a;43:209-23.

Kyriakopoulos CE, Chen YH, Carducci MA et al. Chemohormonal therapy in metastatic hormone-sensitive prostate cancer: long-term survival analysis of the randomized phase III E3805 CHAARTED trial. J Clin Oncol. 2018;36:1080-87.

Lundstrom EA, Rencken RK, van Wyk JH et al. Triptorelin 6-month formulation in the management of patients with locally advanced and metastatic prostate cancer. Clin Drug Investig 2009; 29(12):757-65.

National Health Commission China. Chinese guidelines for diagnosis and treatment of prostate cancer 2018. Chin J Cancer Res. 2019;31:67-83.

Parmar H, Edwards L, Phillips RH et al. Orchiectomy versus long-acting DTrp-6-LHRH in advanced prostatic cancer. Br J Urol 1987;59:248-54.

#### IPSEN GROUP D-CN-52014-237

### CONFIDENTIAL PROTOCOL: FINAL with Amendment 3: Version 4.0, 08 March 2024


| Sponsor | Signa | tory: |
|---------|-------|-------|

PPD 18/03/2024
Date

Medical Development Director

R&D Shanghai Innovation Hub Ipsen (Shanghai)

Unit 01, 15th Floor

No.218, Xujiahui Road

Huangpu District

Shanghai 200001

China

#### Medical Monitor Name and Contact Information:

PPD

Medical Development Director

R&D Shanghai Innovation Hub Ipsen (Shanghai)

Unit 01, 15th Floor

No.218, Xujiahui Road

Huangpu District

Shanghai 200001

China

Telephone: PPD

# dcn52014237v4.0 2024March08\_SponsorSignat ure page

Final Audit Report 2024-03-18

| Created: | 2024-03-18 (Central European Time) PPD |
|------------------------------|----------------------------------------|
| Status: | Signed |
| Transaction ID: | PPD |
| Number of Documents: | 1 |
| Document page count: | 1 |
| Number of supporting files: | 0 |
| Supporting files page count: | 0 |

## "dcn52014237v4.0 2024March08\_SponsorSignature page" History



